| 1 | The Pediatric Artificial Pancreas (PEDAP) trial: A |
|---|----------------------------------------------------|
| 2 | Randomized Controlled Comparison of the Control- |
| 3 | IQ technology Versus Standard of Care in Young |
| 4 | Children in Type 1 Diabetes |

| 5 | <u>Study Sponsor</u> |
|----|--------------------------------------------------------|
| 6 | Marc D. Breton, Ph.D. |
| 7 | University of Virginia |
| 8 | Center for Diabetes Technology |
| 9 | <u>Protocol Chair</u> |
| 10 | R. Paul Wadwa, MD |
| 11 | Barbara Davis Center |
| 12 | University of Colorado |
| 13 | <b>Participating Institutions</b> |
| 14 | University of Virginia, Charlottesville, Virginia |
| 15 | Barbara Davis Center, University of Colorado, Colorado |
| 16 | Stanford University, California |
| 17 | |
| 18 | <b>Coordinating Center</b> |
| 19 | Jaeb Center for Health Research |
| 30 | |
| 20 | |
| 21 | |
| 22 | |
| | N N. 1 44.0 / NICITUO ARO CERO |
| 23 | Version Number: v11.0 / NCT#04796779 |
| 24 | DECEMBER 3 2021 |

| Sponsor Chair / IDE Chair | |
|---|---|
| Name, degree | Marc D. Breton, Ph.D. |
| Institution Name | University of Virginia, Center for Diabetes Technology |
| Protocol Chair/Director | |
| Name, degree | R. Paul Wadwa, MD |
| Institution Name | Barbara Davis Center, University of Colorado |
| JCHR Coordinating Center Director | |
| Name, degree | John Lum, MS |
| Institution Name | Jaeb Center for Health Research |
| Medical Monitor | |
| Name, degree | Roy Beck, M.D., Ph.D. |
| Institution Name | Jaeb Center for Health Research |

| Version<br>Number | Author(s) | Approver | Effective<br>Date | Revision Description |
|---|---|---|---|---|
| 1.0 | R. Paul Wadwa<br>John Lum<br>Roy Beck | R. Paul Wadwa | 23 Nov 2020 | Original protocol |
| 2.0 | John Lum | R. Paul Wadwa | 21 Dec 2020 | Pre-clinical revisions to accommodate requests for changes by IRB and FDA reviewers |
| 3.0 | John Lum | R. Paul Wadwa | 13 Jan 2021 | Pre-clinical revisions to accommodate request by IRB reviewers for changes to framing of extension phase participation |
| 4.0 | John Lum | R. Paul Wadwa | 29 Jan 2021 | Pre-clinical revisions to visit window details in Chapters 5 and 6 to ensure that window definitions are consistent between RCT and Extension period and that associated body text agrees with visit window table text. Initial version used for study. |
| 5.0 | Shannon Hiser, John<br>Lum | R. Paul Wadwa | 7 May 2021 | Addition of inclusion criterion requiring U.S. residency; typo correction in 9.2.4 |
| 6.0 | John Lum | R. Paul Wadwa | 16 Jun 2021 | Addition of SUS Questionnaire, addition of the use of the new version of Control-IQ for the extension phase of the study, updated statistical analyses for the extension phase of the study. |
| 7.0 | John Lum | R. Paul Wadwa | 15 Jul 2021 | Per FDA request, inclusion of all study participants in the 13 week + 3 day call, 14-week call, and 15-week visit |
| 8.0 | John Lum | R. Paul Wadwa | 10 Sep 2021 | Addition of ancillary study during Extension Phase to obtain system performance data during meal/exercise challenges; associated revisions to Stats chapter, plus minor unrelated Stats edits. |
| 9.0 | John Lum | R. Paul Wadwa | 04 Oct 2021 | Revisions to exercise and meal bolus challenges to address FDA requests during IDE review |
| 10.0 | John Lum | R. Paul Wadwa | 26 Oct 2021 | Revisions to exercise and meal bolus challenges to address IRB requests during IRB review |
| 11.0 | John Lum | R. Paul Wadwa | 03 Dec 2021 | Introduction of Extended Use period |

| 31 | CHAPTER 1: BACKGROUND INFORMATION |
|----|----------------------------------------------------------------|
| 32 | 1.1 Introduction |
| 33 | 1.2 Rationale |
| 34 | 1.3 Potential Risks and Benefits of the Investigational Device |
| 35 | 1.3.1 Known Potential Risks |
| 36 | 1.3.1.1 Potential Risks and Benefits of the CLC System |
| 37 | 1.3.1.2 Risk of Hypoglycemia |
| 38 | 1.3.1.3 Risk of Hyperglycemia |
| 39 | 1.3.1.4 Fingerstick Risks |
| 40 | 1.3.1.5 Subcutaneous Catheter Risks (CGM) |
| 41 | 1.3.1.6 Risk of Device Reuse |
| 42 | 1.3.1.7 Questionnaires and Focus Groups |
| 43 | 1.3.1.8 Other Risks |
| 44 | 1.3.2 Known Potential Benefits |
| 45 | 1.3.3 Risk Assessment |
| 46 | 1.4 General Considerations 25 |
| 47 | CHAPTER 2: STUDY ENROLLMENT AND SCREENING |
| 48 | 2.1 Participant Recruitment and Enrollment |
| 49 | 2.1.1 Informed Consent and Authorization Procedures |
| 50 | 2.2 Participant Inclusion Criteria |
| 51 | 2.3 Participant Exclusion Criteria |
| 52 | 2.4 Eligibility Assessment and Baseline Data Collection |
| 53 | 2.5 Historical Information |
| 54 | 2.6 Screening Testing and Procedures 29 |
| 55 | 2.7 Screen Failures |
| 56 | CHAPTER 3: CGM RUN-IN PHASE31 |
| 57 | 3.1 CGM Run-in Phase Overview |
| 58 | 3.2 Initiation of CGM |
| 59 | 3.2.1 CGM Training |
| 60 | 3.3 Blood Glucose and Ketone Testing |
| 61 | 3.4 Assessment of Successful Completion of the Run-in Phase |

| 62 | 3.5 Optimization of Insulin Therapy | 33 |
|----|--------------------------------------------------------------------|----|
| 63 | CHAPTER 4: RANDOMIZATION VISIT | 34 |
| 64 | 4.1 Visit Timing | 34 |
| 65 | 4.1.1 Randomization | 34 |
| 66 | 4.1.2 Baseline HbA1c Determination | 34 |
| 67 | CHAPTER 5: MAIN STUDY PROCEDURES | 35 |
| 68 | 5.1 Visit and Contact Schedule | 35 |
| 69 | 5.2 CGM Initiation and Training | 35 |
| 70 | 5.3 Procedures for the CLC Group | 35 |
| 71 | 5.3.1 Study Pump Training | 35 |
| 72 | 5.3.2 Initiation of Pump by MDI Participants | 36 |
| 73 | 5.3.3 System Use Guidelines | 37 |
| 74 | 5.3.4 Home Use of the Study System | 37 |
| 75 | 5.3.5 Study Device Download | 38 |
| 76 | 5.3.6 3-Day Phone Contact | 38 |
| 77 | 5.3.7 1-Week Phone Contact | 38 |
| 78 | 5.3.8 2-Week Visit | 38 |
| 79 | 5.4 Procedures for the SC Group | 39 |
| 80 | 5.4.1 Study Device Data Download | 39 |
| 81 | 5.4.2 1-Week Phone Contact | 39 |
| 82 | 5.4.3 2-Week Visit | 39 |
| 83 | 5.5 Follow-up Visits and Phone Contacts for Both Groups | 40 |
| 84 | 5.5.1 Visits | 40 |
| 85 | 5.5.2 Phone Contacts | 40 |
| 86 | 5.5.3 Optimization of Insulin Therapy | 40 |
| 87 | 5.5.4 13-Week Visit | 41 |
| 88 | 5.6 Early Termination Visit (If Applicable) | 41 |
| 89 | 5.7 Unscheduled Visits | 41 |
| 90 | CHAPTER 6: EXTENSION PHASE PROCEDURES | 42 |
| 91 | 6.1 Visit and Contact Schedule | 42 |
| 92 | 6.2 Study Pump Initiation | 42 |
| 93 | 6.3 Visits, Videoconferences, and Phone Calls for All Participants | 43 |
| 94 | 6.3.1 13-Week + 3-Day Phone Contact | 43 |

| 95 | 6.3.2 14-Week Phone Contact | 43 |
|---|---|---|
| 96 | 6.3.3 15-Week Visit | 43 |
| 97 | 6.3.4 19-Week Visit | 43 |
| 98 | 6.3.5 23-Week Phone Call | 43 |
| 99 | 6.3.6 26-Week Visit | 43 |
| 100 | 6.3.7 Optimization of Insulin Therapy | 43 |
| 101 | 6.4 Unscheduled Visits | 43 |
| 102 | 6.5 Participant Access to Study Device at Study Closure | 44 |
| 103 | CHAPTER 7: EXTENDED USE PERIOD PROCEDURES | 45 |
| 104 | 7.1 Visit and Contact Schedule | 45 |
| 105 | 7.2 Visits, Videoconferences, and Phone Calls for Participants Re-Initiating Study Pump V | |
| 106 | After a Gap in Use | |
| 107 | 7.2.1 Study Pump Retraining Visit | 45 |
| 108 | 7.2.2 3-Day Phone Contact | |
| 109 | 7.2.3 1-Week Phone Contact | 46 |
| 110 | 7.3 Visits, Videoconferences, and Phone Calls for All Participants | 46 |
| 111 | 7.3.1 13-Week Visit and Subsequent Visits Every 13 Weeks | 46 |
| 112 | 7.3.2 Final Visit | 46 |
| 113 | 7.3.3 Optimization of Insulin Therapy | |
| 114 | 7.4 Unscheduled Visits | 47 |
| 115 | 7.5 Participant Access to Study Device at Study Closure | 47 |
| 116 | CHAPTER 8: STUDY DEVICES | 48 |
| 117 | 8.1 Description of the Investigational Device | 48 |
| 118 | 8.1.1 Insulin Pump | 48 |
| 119 | 8.1.2 Continuous Glucose Monitoring | 48 |
| 120 | 8.1.3 Blood Glucose Meter and Strips | 48 |
| 121 | 8.1.4 Ketone Meter and Strips | 48 |
| 122 | 8.1.5 Study Device Accountability Procedures | 48 |
| 123 | 8.1.6 Blood Ketone Testing | 48 |
| 124 | 8.2 Safety Measures | 48 |
| 125 | 8.2.1 CGM Calibration | 48 |
| 126 | 8.2.2 System Failure | 49 |
| 127 | 8.2.3 Hypoglycemia Threshold Alert and Safety Protocol | 49 |

| 128 | 8.2.4 Hyperglycemia Threshold Alert and Safety Protocol | 49 |
|---|---|---|
| 129 | CHAPTER 9: TESTING PROCEDURES, QUESTIONNAIRES, AND FOCUS GROUPS | 51 |
| 130 | 9.1 Laboratory Testing | 51 |
| 131 | 9.1.1 HbA1c: | 51 |
| 132 | 9.2 Questionnaires | 51 |
| 133 | 9.2.1 PedsQL Diabetes Module – Parent | 51 |
| 134 | 9.2.2 Pediatric Inventory for Parents | 51 |
| 135 | 9.2.3 INSPIRE Survey – Parent | 51 |
| 136 | 9.2.4 Pittsburgh Sleep Quality Index (PSQI) – Parent | 52 |
| 137 | 9.2.5 Hypoglycemia Fear Survey-Parent (HFS-P) | 52 |
| 138 | 9.2.6 Hypoglycemia Confidence Scale | 52 |
| 139 | 9.2.7 System Usability Scale (SUS) | 52 |
| 140 | 9.3 Focus Groups | 53 |
| 141 | CHAPTER 10: UNANTICIPATED PROBLEM, ADVERSE EVENT, AND DEVICE ISSUES REPORTING. | 54 |
| 142 | 10.1 Unanticipated Problems | 54 |
| 143 | 10.2 Adverse Events | 54 |
| 144 | 10.2.1 Definitions | 54 |
| 145 | 10.2.2 Reportable Adverse Events | 55 |
| 146 | 10.2.3 Hypoglycemic Events | 56 |
| 147 | 10.2.4 Hyperglycemic/Ketotic Events | 56 |
| 148 | 10.2.5 Relationship of Adverse Event to Study Device | 57 |
| 149 | 10.2.6 Severity (Intensity) of Adverse Events | 57 |
| 150 | 10.2.7 Expectedness | 58 |
| 151 | 10.2.8 Coding of Adverse Events | 58 |
| 152 | 10.2.9 Outcome of Adverse Events | 58 |
| 153 | 10.3 Reportable Device Issues | 59 |
| 154 | 10.4 Timing of Event Reporting | 59 |
| 155 | 10.5 Safety Oversight | 60 |
| 156 | 10.6 Stopping Criteria | 60 |
| 157 | 10.6.1 Participant Discontinuation of Study Device | 60 |
| 158 | 10.6.2 Criteria for Suspending or Stopping Overall Study | 61 |
| 159 | CHAPTER 11: MISCELLANEOUS CONSIDERATIONS | |
| 160 | 11.1 Drugs Used as Part of the Protocol | 62 |

| 161 | 11.2 Collection of Medical Conditions and Medications | 62 |
|---|---|---|
| 162 | 11.3 Prohibited Medications, Devices, Treatments, and Procedures | 62 |
| 163 | 11.4 Precautionary Medications, Treatments, and Procedures | 62 |
| 164 | 11.5 Prophylactic Medications, Treatments, and Procedures | 62 |
| 165 | 11.6 Rescue Medications, Treatments, and Procedures | 63 |
| 166 | 11.7 Participant Compensation | 63 |
| 167 | 11.8 Participant Withdrawal | 63 |
| 168 | 11.9 Confidentiality | 63 |
| 169 | CHAPTER 12: STATISTICAL CONSIDERATION | 64 |
| 170 | 12.1 Statistical and Analytical Plans | 64 |
| 171 | 12.2 Statistical Hypotheses | 64 |
| 172 | 12.3 Sample Size | 64 |
| 173 | 12.4 Efficacy Outcome Measures | 65 |
| 174 | 12.4.1 Primary Efficacy Endpoint | 65 |
| 175 | 12.4.2 Secondary Efficacy Endpoints | 65 |
| 176 | 12.4.2.1 Secondary Efficacy Endpoints Included in Hierarchical Analysis | 65 |
| 177 | 12.4.2.2 Other Secondary Efficacy Endpoints | 65 |
| 178 | 12.4.3 CGM Metrics Calculations | 66 |
| 179 | 12.5 Analysis Datasets and Sensitivity Analyses | 67 |
| 180 | 12.5.1 Per Protocol Analyses | 67 |
| 181 | 12.5.2 Other Sensitivity Analyses | 67 |
| 182 | 12.6 Analysis of the Primary Efficacy Endpoint | 68 |
| 183 | 12.7 Analysis of the Secondary Endpoints | 68 |
| 184 | 12.7.1 Hierarchical Analyses | 68 |
| 185 | 12.7.2 Other Endpoint Analyses | 69 |
| 186 | 12.8 Safety Analyses | 70 |
| 187 | 12.9 Intervention Adherence | 71 |
| 188 | 12.10 Protocol Adherence and Retention | 71 |
| 189 | 12.11 Baseline Descriptive Statistics | 71 |
| 190 | 12.12 Device Issues | 72 |
| 191 | 12.13 Planned Interim Analyses | 72 |
| 192 | 12.14 Subgroup Analyses | 72 |
| 193 | 12.15 Multiple Comparison/Multiplicity | 73 |

| 194 | 12.16 Exploratory Analyses | 73 |
|---|---|---|
| 195 | 12.17 Extension Phase | 74 |
| 196 | 12.17.1 Exclusion of Ancillary Study Data | 75 |
| 197 | 12.18 Extended Use Period. | 75 |
| 198 | CHAPTER 13: DATA COLLECTION AND MONITORING | 76 |
| 199 | 13.1 Case Report Forms and Device Data | 76 |
| 200 | 13.2 Study Records Retention | 76 |
| 201 | 13.3 Quality Assurance and Monitoring | 76 |
| 202 | 13.4 Protocol Deviations | 77 |
| 203 | CHAPTER 14: ETHICS/PROTECTION OF HUMAN PARTICIPANTS | 78 |
| 204 | 14.1 Ethical Standard | 78 |
| 205 | 14.2 Institutional Review Boards | 78 |
| 206 | 14.3 Informed Consent Process | 78 |
| 207 | 14.3.1 Consent Procedures and Documentation | 78 |
| 208 | 14.3.2 Participant and Data Confidentiality | 78 |
| 209<br>210 | CHAPTER 15: ANCILLARY STUDY TO TEST CONTROL-IQ SYSTEM WITH MEAL BOLUS A | |
| 211 | 15.1 Objective | |
| 212 | 15.2 Sample Size | |
| 213 | 15.3 Eligibility Criteria | |
| 214 | 15.4 Study Procedures | 80 |
| 215 | 15.5 Outcomes and Analysis Plan | 82 |
| 216 | Safety Monitoring | 83 |
| 217 | CHAPTER 16: REFERENCES | 84 |

| ABBREVIATION | DEFINITION |
|--------------|-------------------------------------------|
| AP | Artificial Pancreas |
| BG | Blood Glucose |
| BT/BTLE | Bluetooth, Bluetooth low energy |
| CRF | Case Report Form |
| CGM | Continuous Glucose Monitoring System |
| CLC | Closed-Loop Control |
| CSII | Continuous Subcutaneous Insulin Injection |
| CTR | Control-to-Range |
| DiAs | Diabetes Assistant |
| DKA | Diabetic Ketoacidosis |
| EC | European Commission |
| FDA | Food and Drug Administration |
| GCP | Good Clinical Practice |
| HbA1c | Hemoglobin A1c |
| ID | Identification |
| iDCL | International Diabetes Closed Loop |
| IDE | Investigational Device Exemption |
| IOB | Insulin-on-Board |
| IQR | Interquartile Range |
| JDRF | Juvenile Diabetes Research Foundation |
| LGS | Low Glucose Suspend |
| PLGS | Predictive Low Glucose Suspend |
| POC | Point-of-Care |
| QA | Quality Assurance |
| QC | Quality Control |
| RBM | Risk-Based Monitoring |
| RCT | Randomized Control Trial |
| SC | Standard of Care group |
| SD | Standard Deviation |
| TDD | Total Daily Dose |
| UI | User Interface |

# **Signature Page**

Translation of the UVA Advanced Automated Insulin Delivery
Systems to Clinical Care in Young Children: Glycemic Control,
Regulatory Acceptance, and Optimization of Day to Day Use

226 **Protocol Identifying Number: PEDAP** 

227 IND/IDE Sponsor: University of Virginia

Version Number: 11.0

229 **03 DEC 2021** 

| Protocol Chair | |
|---|---|
| Name, Institution | R. Paul Wadwa, M.D. / University of Colorado – Barbara Davis Center |
| Signature/Date | |
| Sponsor (IDE Holder) | |
| Name/Institution | Marc D. Breton, Ph.D. / University of Virginia |
| Signature/Date | |
| <b>Coordinating Center Director</b> | |
| Name, Institution | John Lum, MS / Jaeb Center for Health Research |
| Signature/Date | |
| Medical Monitor | |
| Name, Institution | Roy Beck, MD, Ph.D. / Jaeb Center for Health Research |
| Signature/Date | |

| 230 | CLINICAL CENTER PRINCIPAL INVESTIGATOR STATEMENT OF | | | | |
|---|---|---|---|---|---|
| 231 | COMPLIANCE | | | | |
| 232<br>233<br>234 | Protocol Title: The Pediatric Artificial Pancreas (PEDAP) trial: Comparison of the Control-IQ technology Versus Standard of Type 1 Diabetes | | | | |
| 235 | Protocol Version/Date: 11.0 / 03 DEC 2021 | | | | |
| 236<br>237<br>238<br>239<br>240<br>241 | I have read the protocol specified above. In my formal capacity as Investigator, my duties include ensuring the safety of the study part supervision and providing the Jaeb Center for Health Research, wit information, as outlined in the protocol. It is understood that all instudy will be held strictly confidential and that this confidentiality is study staff at this clinical center. | cicipants en<br>h complete<br>Formation p | rolled un<br>and time<br>ertaining | nder r<br>ely<br>g to tl | ny<br>ne |
| 242<br>243<br>244<br>245 | This trial will be carried out in accordance with ICH E6 Good Clin required by the following: United States (US) Code of Federal Reg clinical studies (45 CFR Part 46, 21 CFR Part 50, 21 CFR Part 56, CFR Part 812). | ulations (C | FR) app | licabl | e to |
| 246<br>247<br>248<br>249 | As the Principal Investigator, I will assure that no deviation from, of will take place without prior agreement from the sponsor and document institutional Review Board (IRB), or other approved Ethics Committo eliminate an immediate hazard(s) to the trial participants. | nented app | roval fro | om th | e |
| 250<br>251<br>252<br>253 | All key personnel (all individuals responsible for the design and co<br>completed Human Participants Protection Training and Good Clini<br>Further, I agree to ensure that all staff members involved in the con<br>informed about their obligations in meeting the above commitment | cal Practice duct of this | Trainin | ıg. | |
| 254<br>255 | Investigator's Signature | Date: | // | / _ | уууу |
| 256 | Investigator's Name: | | | | |
| 257 | Clinical Center Name/Number: | | | | |

## PROTOCOL SUMMARY

| PARTICIPANT AREA | DESCRIPTION |
|---|---|
| Title | The Pediatric Artificial Pancreas (PEDAP) trial: A Randomized<br>Controlled Comparison of the Control-IQ technology Versus Standard<br>Care in Young Children in Type 1 Diabetes |
| Précis | A randomized controlled trial of at-home closed loop system vs. standard care (defined as either multiple daily injections of insulin [MDI] or use of an insulin pump without hybrid closed-loop control capabilities [low-glucose suspend or predictive low-glucose suspend functionality is permitted]) in youth age 2 to <6 years old. |
| Investigational Device | t:slim X2 with Control-IQ and Dexcom G6 system |
| Objectives | The objective of the study is to assess efficacy, quality of life, and safety of a closed loop control (CLC) system (t:slim X2 with Control-IQ Technology) in a randomized controlled trial with partial crossover. |
| Study Design | First phase: a 13-week parallel group randomized clinical trial with 2:1 randomization to intervention with the closed loop system vs. standard care (SC); Second Phase: following the RCT, a 13-week period where the Standard Care (SC) group will transition to use CLC and the experimental arm will extend the use of CLC for the same period. After 26 weeks, participants may continue using CLC for an additional Extended Use period. A subset of participants will be invited to join an optional exercise/meal challenge ancillary study. |
| <b>Number of Clinical Centers</b> | ~3 US clinical centers |
| Endpoints | Efficacy The primary outcome for the RCT is time in target range 70-180 mg/dL (TIR) measured by CGM in CLC group vs. SC group over 13 weeks The primary outcome for the extension phase assessed separately for each treatment group is change in TIR comparing extension phase with RCT phase. Ouality of Life Patient-reported outcome questionnaires will be completed. Safety The key safety outcomes are severe hypoglycemia and ketoacidosis. |
| Population | <ol> <li>Inclusion Criteria</li> <li>Clinical diagnosis, based on investigator assessment, of type 1 diabetes for at least 6 months and using insulin for at least 6 months</li> <li>Familiarity and use of a carbohydrate ratio for meal boluses.</li> <li>Age ≥2 and &lt;6 years old</li> <li>Living with one or more parent/legal guardian knowledgeable about emergency procedures for severe hypoglycemia and able to contact emergency services and study staff.</li> <li>Investigator has confidence that the parent can successfully operate all study devices and is capable of adhering to the protocol</li> <li>Willingness to switch to lispro (Humalog) or aspart (Novolog) if not using already, and to use no other insulin besides lispro (Humalog) or aspart (Novolog) during the study for participants using a study-provided Tandem pump during the study.</li> <li>Total daily insulin dose (TDD) at least 5 U/day</li> <li>Body weight at least 20 lbs</li> </ol> |

| PARTICIPANT AREA | DESCRIPTION |
|---|---|
| | <ol> <li>Willingness not to start any new non-insulin glucose-lowering agent during the course of the trial</li> <li>Participant and parent(s)/guardian(s) willingness to participate in all training sessions as directed by study staff.</li> <li>Parent/guardian proficient in reading and writing English</li> <li>Live in the United States, with no plans to move outside the United States during the study period</li> </ol> |
| | <ol> <li>Exclusion Criteria</li> <li>Concurrent use of any non-insulin glucose-lowering agent (including GLP-1 agonists, Symlin, DPP-4 inhibitors, SGLT-2 inhibitors, sulfonylureas).</li> <li>Hemophilia or any other bleeding disorder</li> <li>History of &gt;1 severe hypoglycemic event with seizure or loss of consciousness in the last 3 months</li> <li>History of &gt;1 DKA event in the last 6 months not related to illness, infusion set failure, or initial diagnosis</li> <li>History of chronic renal disease or currently on hemodialysis</li> <li>History of adrenal insufficiency</li> <li>Hypothyroidism that is not adequately treated</li> <li>Use of oral or injectable steroids within the last 8 weeks</li> <li>Known, ongoing adhesive intolerance</li> <li>Plans to receive blood transfusions or erythropoietin injections during the course of the study</li> <li>A condition, which in the opinion of the investigator or designee, would put the participant or study at risk</li> <li>Currently using any closed-loop system, or using an insulin pump that is incompatible with use of the study CGM</li> <li>Participation in another pharmaceutical or device trial at the time of enrollment or during the study</li> <li>Employed by, or having immediate family members employed by Tandem Diabetes Care, Inc., or having a direct supervisor at place of employment who is also directly involved in conducting the clinical trial (as a study investigator, coordinator, etc.); or having a first-degree relative who is directly involved in conducting the clinical trial</li> </ol> |
| Sample Size | Up to 150 screened participants with the goal of randomizing 102 participants. |
| Treatment Groups | Intervention Group: t:slim X2 with Control-IQ Technology and Study CGM. Control Group: Standard care (SC) - defined as either multiple daily injections of insulin (MDI) or use of an insulin pump without hybrid closed-loop control capabilities (low-glucose suspend or predictive low-glucose suspend functionality is permitted) in conjunction with study CGM |
| | All participants will be offered to extend the study for an additional 13 weeks, with the SC group switching to the t:slim X2 with Control-IQ System after the 13-week RCT period. After 26 weeks, participants may continue using CLC for an additional Extended Use period. |
| Participant Duration | ~26-32 weeks for RCT and Extension Phase, depending on duration of run-in phase; up to an additional ~7 months in Extended Use period |
| Protocol Overview/Synopsis | After consent is signed, eligibility will be assessed. Eligible participants not currently using an insulin pump and Dexcom G5 or Dexcom G6 CGM with minimum data requirements will initiate a run-in phase of 2 to 6 weeks that will be customized based on whether the participant is already |

| PARTICIPANT AREA | DESCRIPTION |
|---|---|
| | a CGM user. Participants who skip or successfully complete the run-in will be randomly assigned 2:1 to an intervention using Tandem t:slim X2 with Control-IQ Technology or the standard care control group using existing insulin therapy in conjunction with study CGM. All participants will continue their participation by using the t:slim X2 with Control-IQ system in an Extension Phase. [Figure 1] After 26 weeks, participants may continue using CLC for an additional Extended Use period through no later than July 31, 2022. A subset of participants will complete an optional exercise/meal challenge ancillary study. |



Figure 1: Study Design: Participants Randomized 2:1 Control-IQ Control (CLC) vs. Standard Care (SC) Groups. Extension phase with partial crossover of SC Group switching to use Control-IQ. Subsequent Extended Use period through no later than July 31, 2022.

262

263264



<sup>\*</sup>Current use of Dexcom G5 or G6 CGM with readings captured on at least 11 out of the previous 14 days

Figure 2: Overview of Study Design



Figure 3: Schematic of Study Design (Post-Randomization through 26 Weeks)



<sup>\*</sup> Final Visit to occur no later than July 31, 2022

Figure 4: Schematic of Study Design (Extended Use Period)

277

| VC/V | | | | | | | | | 3d | 14w | 15w | 19w | 23w | 26w |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | VC/V | VC/V | VC/<br>P | P | VC/V | VC/<br>V | P | VC/<br>V | VC/<br>P | P | VC/<br>V | VC/<br>V | P | VC/<br>V |
| Screen/<br>Enroll | Run-in | Rand | | | | | | | | | | | | |
| X | X | X | | | | | | | | | | | | |
| | | X | | | | | | X | | | | | | X |
| X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| X | | | | | | | | X | | | | | | X |
| | X X X | Enroll Run-in X X X X X X X X | Enroll Run-in Rand X X X X X X X X X X X X | Run-in Rand | Enroll Run-in Rand X X X X X X X X X X X X X X X | Run-in Rand | Enroll Run-in Rand X X X X X X X X X X X X X X X X X X X X | Enroll Run-in Rand X X X X X X X X X X X X X X X X X X X X | Enroll Run-in Rand X X X X X X X X X X X X X X X X X X X X X X X X X | Enroll Run-in Rand X X X X X X X X X X X X X X X X X X X X X X X X X | Enroll Run-in Rand X X X X X X X X X X X X X X X X X X X X X X X X X X X X X | Enroll Run-in Rand X X X X X X X X X X X X X X X X X | Enroll Run-in Rand X X X X X X X X X X X X X X X X X | Enroll Run-in Rand Image: Control of the control of |

<sup>&</sup>lt;sup>1</sup> Only for participants on MDI at enrollment assigned to the CLC group

276 Table 1. Schedule of Study Visits and Procedures (through 26-Week Visit)

| _ | | | | | | 2=0 |
|---|---|---|---|---|---|---|
| Days/Weeks after<br>26-Week Visit => | $0^2$ | $3d^2$ | 1w <sup>2</sup> | 13w | 26w, 39w,<br>etc. | Final<br>Visit |
| Visit (V),<br>Videoconference (VC),<br>or Phone (P) | VC/V | VC/<br>P | VC/<br>P | VC/V | VC/V | VC/V |
| Eligibility Assessment <sup>1,2</sup> | X | | | | | |
| Study Pump Retraining <sup>2</sup> | X | | | | | |
| HbA1c (Central lab) | | | | X | X | |
| Device Data download(s) | | X | X | X | X | X |
| Review diabetes<br>management and AEs | | X | X | X | X | X |

<sup>1</sup> Participants are eligible to initiate Extended Use period if they completed the 26-Week Visit within the prior 4 months

<sup>2</sup> Only for participants who had a gap between the 26-Week Visit and the initiation of the Extended Use period during which they stopped use of the study pump and reverted to MDI or personal pump insulin therapy

Table 2. Schedule of Study Visits and Procedures (Extended Use Period)

## **Chapter 1: Background Information**

### 1.1 Introduction

294

295

302

- The Tandem X2 insulin pump with Control-IQ Technology is a third-generation closed-loop
- control (CLC) system retaining the same control algorithm that was initially tested by UVA's DiAs
- 298 system and then implemented in the inControl system (TypeZero Technologies, Inc.).
- 299 The system has received FDA approval for use in individuals ≥6 years old following a pair of
- 300 pivotal trials that demonstrated the system's safety and efficacy, first in participants ≥14 years old
- 301 (1) and then subsequently in participants  $\geq 6$  years old (2).

## Closed-Loop Control System

- The Closed-Loop Control System contained in t-slim X2 with Control-IQ Technology is described
- in Master File MAF-2032/A008. Control-IQ Technology is derived from inControl previously
- described in IDE# G160097, G160181, G150240 and G140169/S010. The CLC is an "artificial
- pancreas" (AP) application that uses advanced closed loop control algorithms to automatically
- manage blood glucose levels for people with Type 1 Diabetes. The system modulates insulin to
- 308 keep blood glucose in a targeted range. The system components include the t:slim X2 with
- 309 Control-IQ Technology and the Dexcom CGM G6.



310311

Figure 5. t:slim X2 with Control-IQ and Dexcom G6 system

## **1.2 Rationale**

- The objective of this randomized clinical trial is to assess the efficacy and safety of the Control-
- 314 IQ closed loop system over a 13-week period compared with standard care. In addition, the data
- from this trial may be used for subsequent regulatory submissions for this system in the age group
- 316 studied.
- The extension phase will allow for additional exposure time to the Tandem t:slim X2 with Control-
- 318 IQ Technology and evaluation of the SC arm after crossing over to use Control-IQ for a 13-week
- 319 period.

## 320 1.3 Potential Risks and Benefits of the Investigational Device

- Risks and Benefits are detailed below. Loss of confidentiality is a potential risk; however, data are
- handled to minimize this risk. Hypoglycemia, hyperglycemia and ketone formation are always a
- risk in participants with type 1 diabetes and participants will be monitored for these events.

## 1.3.1 Known Potential Risks

324

## 325 1.3.1.1 Potential Risks and Benefits of the CLC System

- Even though the study system has been tested prior to this study, there is still a risk that parts of
- 327 the system may not function properly. The following are possible reasons the system may deliver
- 328 too much insulin or incorrectly stop insulin delivery:
- CGM sensor reads higher or lower than the actual glucose level which increases risk for hypoglycemia and hyperglycemia with automated insulin delivery system;
- Device malfunctions that could produce a suspension of insulin delivery or over delivery of insulin.

## 333 1.3.1.2 Risk of Hypoglycemia

- As with any person having type 1 diabetes and using insulin, there is always a risk of having a low
- blood sugar (hypoglycemia). The frequency of hypoglycemia should be no more and possibly less
- than it would be as part of daily living. Symptoms of hypoglycemia can include sweating,
- 337 jitteriness, and not feeling well. Just as at home, there is the possibility of fainting or seizures
- 338 (convulsions) and that for a few days the participant may not be as aware of symptoms of
- 339 hypoglycemia. A CGM functioning poorly and significantly over-reading glucose values could
- lead to inappropriate insulin delivery.

## 341 1.3.1.3 Risk of Hyperglycemia

- 342 Hyperglycemia and ketonemia could occur if insulin delivery is attenuated or suspended for an
- extended period or if the pump or infusion set is not working properly. A CGM functioning poorly
- and significantly under-reading glucose values could lead to inappropriate suspension of insulin
- 345 delivery.

## 346 1.3.1.4 Fingerstick Risks

- 347 At various times several drops of blood will be removed by fingerstick. This is a standard method
- used to obtain blood for routine hospital laboratory tests. Pain is common at the time of lancing.
- In about 1 in 10 cases, a small amount of bleeding under the skin will produce a bruise. A small
- scar may persist for several weeks. The risk of local infection is less than 1 in 1000. This should
- not be a significant contributor to risks in this study as fingersticks are part of the usual care for
- people with diabetes.

## 353 1.3.1.5 Subcutaneous Catheter Risks (CGM)

- Participants using the CGM will be at low risk for developing a local skin infection at the site of
- 355 the sensor needle placement. If a catheter is left under the skin for more than 24 hours, it is possible

- 356 to get an infection where it goes into the skin, with swelling, redness and pain. There may be
- 357 bleeding where the catheter is put in and bleeding under the skin causes a bruise (1 in 10 risk).
- 358 Study staff should verbally alert the participant that on rare occasions, the CGM may break and
- leave a small portion of the sensor under the skin that may cause redness, swelling or pain at the
- 360 insertion site. The participant should be further instructed to notify the study coordinator
- immediately if this occurs.

379

386

## 1.3.1.6 Risk of Device Reuse

- 363 The study CGM system is labeled for single use only. The sensor (the component of the system
- that enters the skin) will be single use only. The receiver, if used, is a hand-held device. The
- transmitter and receiver may be reused during the study after cleaning the device using a hospital-
- approved cleaning procedure. The transmitter is attached to the sensor but does not enter the skin.
- Participants will be informed that FDA or relevant national authorities have approved these devices
- for single use and that by using them among multiple patients, bloodborne pathogens (i.e. Hepatitis
- B) may be spread through the use of multiple users.
- 370 The study insulin pump is labeled for single-patient use. During the study, this device may be
- 371 reused after cleaning adhering to a hospital-approved cleaning procedure. All infusion set
- equipment will be single patient use only (infusion set insertion kits, tubing, cartridges etc.)
- Participants will be informed that FDA or relevant national authorities typically approve the insulin
- pump device for single use and that by using them among multiple patients, bloodborne pathogens
- 375 (i.e. Hepatitis B) may be spread through the use of multiple users.
- 376 The study blood glucose meter and blood ketone meter are labeled for single-patient use.
- During the study, only one person can use each device as there are rare risks that bloodborne
- pathogens (i.e. Hepatitis B) may be spread through the use of multiple users.

## 1.3.1.7 Questionnaires and Focus Groups

- 380 As part of the study, parents of participants will complete questionnaires which include questions
- 381 about their private attitudes, feelings and behavior related to the investigational equipment as well
- as managing diabetes. Parents may also participate in a focus group session to explore their
- feelings about using the closed-loop system. It is possible that some people may find these
- 384 questionnaires or focus groups to be mildly upsetting. Similar questionnaires and focus groups
- have been used in previous research and these types of reactions have been uncommon.

## 1.3.1.8 Other Risks

- 387 Some participants may develop skin irritation or allergic reactions to the adhesives used to secure
- the CGM, or to secure the insulin infusion sets for the continuous subcutaneous insulin infusion.
- 389 If these reactions occur, different adhesives or "under-taping" (such as with IV 3000, Tegaderm,
- 390 etc.) will be tried, sites will be rotated frequently, and a mild topical steroid cream or other
- medication may be required.
- Whenever the skin is broken there is the possibility of an infection. The CGM and pump infusion
- 393 sites are inserted under the skin. It is possible that any part that is inserted under the skin may

- 394 cause an infection. These occur very infrequently, but, if an infection was to occur, oral and/or
- 395 topical antibiotics can be used. The risk of skin problems could be greater if you use a sensor for
- longer than it is supposed to be used. Therefore, participants (and parents) will be carefully
- instructed about proper use of the sensor.
- Data downloaded from the CGM, pump, and the home glucose and ketone meter will be collected
- 399 for the study as measures of diabetes self-management behaviors. Some people
- 400 may be uncomfortable with the researchers' having such detailed information about their daily
- 401 diabetes habits.

423

## 1.3.2 Known Potential Benefits

- 403 One purpose of this research is to reduce the frequency of hypoglycemia and severe hypoglycemic
- events. Hypoglycemia is the number one fear of many individuals and families with someone who
- has type 1 diabetes and this fear often prevents optimal glycemic control.
- 406 It is expected that this protocol will yield increased knowledge about using an automated
- 407 closed-loop system to control the glucose level and is intended to develop data to support future
- device approval in the age group studied. The individual participant may not benefit from study
- 409 participation.

## 410 **1.3.3 Risk Assessment**

- 411 Based on the facts that (1) children with diabetes experience mild hypoglycemia and
- 412 hyperglycemia frequently as a consequence of the disease and its management, (2) the study
- 413 intervention involves periodic automated insulin dosing that may reduce the likelihood of
- 414 hypoglycemia, and periodic automated attenuation of insulin delivery that may reduce the
- 415 likelihood of hyperglycemia, (3) if any, hypo and/or hyperglycemia occur, mitigations are in place,
- and have been tested in prior studies using the investigational device system in the home setting,
- 417 that limit the likelihood of excessive insulin dosing or prolonged withdrawal of insulin, and (4)
- 418 rapid reversal of hypoglycemia and hyperglycemia can be achieved, it is the assessment of the
- investigators that this protocol falls under DHHS 45 CFR 46.405 and 21 CFR 50.52 as a clinical
- 420 investigation involving greater than minimal risk but presenting the prospect of direct benefit to
- 421 individual subjects. In addition, it is the belief of the investigators that this study also presents
- prospect of general benefit to others with diabetes.

#### 1.4 General Considerations

- The study is being conducted in compliance with the policies described in the study policies
- document, with the ethical principles that have their origin in the Declaration of Helsinki, with the
- 426 protocol described herein, and with the standards of Good Clinical Practice (GCP).
- There is no restriction on the number of participants to be enrolled by each clinical center toward
- 428 the overall recruitment goal.
- The protocol is considered a significant risk device study, due to the fact that the closed loop
- 430 system is experimental in the population under study. Therefore, an investigational device

| 431<br>432 | exemption (IDE) from the U.S. Food and Drug Administration (FDA) is required to conduct the study. |
|---|---|

## **Chapter 2: Study Enrollment and Screening**

#### 2.1 Participant Recruitment and Enrollment 434 435 Enrollment will proceed with the goal of having 102 participants randomized. A maximum of 150 436 individuals may be enrolled into screening for the study in order to achieve this goal. 437 Study participants will be recruited at ~3 clinical centers in the United States without regard to 438 gender, race, or ethnicity. There is no restriction on the number of participants to be enrolled by 439 each clinical center toward the overall recruitment goal. 440 The study team will make every effort to have the following minimum numbers of participants 441 complete the trial in the specified subgroups at the time of enrollment: 442 • Approximately two-thirds of the participants with most recent available HbA1c $\geq 7.5\%$ 443 • Approximately 30 participants in the age range >24 months to <48 months 444 • At least 20% of participants who are on multiple daily injections (MDI) rather than pump 445 2.1.1 Informed Consent and Authorization Procedures 446 Potential eligibility may be assessed as part of a routine-care examination. Before completing any 447 procedures or collecting any data that are not part of usual care, electronic informed consent will be obtained. 448 449 A parent/legal guardian (referred to subsequently as "parent") will be provided with the Informed 450 Consent Form to read and will be given the opportunity to ask questions either via 451 phone/videoconference or by mail or email. If the parent and child are interested in the study, the 452 investigator will schedule a virtual or in-person visit to discuss study, and if the parent and child 453 agree to participate, the Informed Consent Form will be electronically signed through the JCHR 454 website. A copy of the electronically signed consent form can be printed by the parent and another 455 copy will be printed by the site to add to the participant's study record. 456 As part of the informed consent process, the parent will be asked to sign an authorization for release 457 of personal information. This may be done electronically with the consent, or on paper if the site 458 requires their own process. The investigator, or his or her designee, will review the study-specific 459 information that will be collected and to whom that information will be disclosed. After speaking 460 with the parent, questions will be answered about the details regarding authorization. 461 A participant is considered enrolled when the informed consent form has been electronically 462 signed and HIPAA authorization has been provided.

Individuals must meet all of the following inclusion criteria in order to be eligible to participate in

2.2 Participant Inclusion Criteria

463

464

465

the study.

- 1. Clinical diagnosis, based on investigator assessment, of type 1 diabetes for at least 6 months and using insulin for at least 6 months
- 468 2. Familiarity and use of a carbohydrate ratio for meal boluses.
- 469 3. Age  $\geq 2$  and  $\leq 6$  years old
- 4. Living with one or more parent/legal guardian knowledgeable about emergency procedures for severe hypoglycemia and able to contact emergency services and study staff.
- 5. Investigator has confidence that the parent can successfully operate all study devices and is capable of adhering to the protocol
- 6. Willingness to switch to lispro (Humalog) or aspart (Novolog) if not using already, and to use no other insulin besides lispro (Humalog) or aspart (Novolog) during the study for participants using a study-provided Tandem pump during the study.
- Study will not be providing insulin; therefore, participants will need to have access to either lispro or aspart
- 7. Total daily insulin dose (TDD) at least 5 U/day
- 480 8. Body weight at least 20 lbs
- 9. Willingness not to start any new non-insulin glucose-lowering agent during the course of the trial (see section 2.3)
- 483 10. Participant and parent(s)/guardian(s) willingness to participate in all training sessions as directed by study staff.
- 485 11. Parent/guardian proficient in reading and writing English
- 12. Live in the United States, with no plans to move outside the United States during the studyperiod

## 488 **2.3 Participant Exclusion Criteria**

- Individuals meeting any of the following exclusion criteria at baseline will be excluded from study participation.
- 1. Concurrent use of any non-insulin glucose-lowering agent (including GLP-1 agonists, Symlin, DPP-4 inhibitors, SGLT-2 inhibitors, sulfonylureas).
- 493 2. Hemophilia or any other bleeding disorder
- 3. History of >1 severe hypoglycemic event with seizure or loss of consciousness in the last 3 months
- 496 4. History of >1 DKA event in the last 6 months not related to illness, infusion set failure, or initial diagnosis
- 498 5. History of chronic renal disease or currently on hemodialysis
- 499 6. History of adrenal insufficiency
- 7. Hypothyroidism that is not adequately treated

- 8. Use of oral or injectable steroids within the last 8 weeks
- 502 9. Known, ongoing adhesive intolerance
- 503 10. Plans to receive blood transfusions or erythropoietin injections during the course of the study
- 11. A condition, which in the opinion of the investigator or designee, would put the participant or study at risk (specified in the study procedure manual); the investigator will take into account the participant's HbA1c level, compliance with current diabetes management, and prior acute
- 507 diabetic complications
- 508 12. Currently using any closed-loop system, or using an insulin pump that is incompatible with use of the study CGM
- 510 13. Participation in another pharmaceutical or device trial at the time of enrollment or during the study
- 512 14. Employed by, or having immediate family members employed by Tandem Diabetes Care, Inc.,
- or having a direct supervisor at place of employment who is also directly involved in
- 514 conducting the clinical trial (as a study investigator, coordinator, etc.); or having a first-degree
- relative who is directly involved in conducting the clinical trial

## **2.4 Eligibility Assessment and Baseline Data Collection**

- Potential participants will be evaluated for study eligibility through the elicitation of a medical
- 518 history and local laboratory testing as needed in the judgment of the investigator (as part of usual
- 519 care).

530

- The screening visit and subsequent scheduled study visits may be conducted virtually via
- videoconference at the discretion of the study investigator, for example due to institutional
- restrictions or the participant or investigator's preference for a remote visit. Study staff will
- discuss the feasibility of conducting virtual visits with each participant and provide support as
- needed to ensure adequate access. The screening visit must be completed within 28 days of
- 525 participant enrollment.

## 526 **2.5 Historical Information**

- A history will be elicited from the parent and extracted from available medical records with
- respect to the participant's diabetes history, current diabetes management, other past and current
- medical problems, past and current medications, and drug allergies.

## 2.6 Screening Testing and Procedures

- At the Screening Visit the following procedures will be performed:
- Informed consent process
- Assessment of eligibility
- Contact information (retained at the clinical center and not entered into study database)
- Demographics (date of birth, sex, race and ethnicity)

| 536 | Measurement of height/weight |
|---|---|
| 537<br>538<br>539 | <ul> <li>If the visit is conducted virtually, a verbal report of the participant's weight and<br/>verbal report of height will be acceptable. A scale will be provided for<br/>participants who do not already have a scale at home.</li> </ul> |
| 540 | • Determination of most recent HbA1c level from medical records or verbal report |
| 541<br>542 | • Participants' parents will complete a set of baseline questionnaires, described in section 9.2. |
| 543 | 2.7 Screen Failures |
| 544<br>545 | Individuals who do not initially meet study eligibility requirements may be rescreened at a later date per investigator discretion. |

# **Chapter 3: CGM Run-In Phase**

| <ul><li>548</li><li>549</li><li>550</li></ul> | This phase must begin (supplies shipped) within 3 days of completion of the Screening visit. The purpose of this CGM run-in phase is to 1) assess compliance with study procedures and 2) to introduce the study CGM to study participants without current use of a Dexcom CGM. |
|---|---|
| 551<br>552<br>553<br>554<br>555 | Participants who currently use a Dexcom G5 or G6 with CGM data captured on at least 11 out of the previous 14 days prior to the time of enrollment can skip the run-in phase. Participants who do not currently use a Dexcom G5 or G6 CGM, or who do use that CGM but have readings captured on fewer than 11 out of the previous 14 days prior to time of enrollment, will be required to participate in the CGM run-in phase. |
| 556<br>557 | Participants and their parent(s) will receive training on the study CGM as detailed below. This will be an unblinded use of the study CGM. |
| 558 | 3.2 Initiation of CGM |
| 559<br>560 | Study CGM supplies will be provided to the participant either in-person at the clinic, or via delivery by other means (personal delivery, overnight shipment, etc.). |
| 561<br>562<br>563 | Once the supplies have been received, the participant and parent will be instructed to use the study CGM on a daily basis. Participants using a personal CGM prior to the study will discontinue the personal CGM beginning in this period. |
| 564 | 3.2.1 CGM Training |
| 565<br>566<br>567<br>568<br>569 | CGM training (in-person or via videoconference) will be provided by a qualified trainer to participants not currently using a personal CGM identical to the study CGM as to how to use it in real-time to make management decisions and how to review the data after an upload for retrospective review. The participating child will participate in training sessions to the degree judged appropriate by the parent and trainer. CGM training will include: |
| 570<br>571 | • Instruction on how to insert the sensor and transmitter, including observation/supervision of placement of a sensor |
| 572 | • Instruction on how to calibrate the CGM unit, if needed |
| 573<br>574<br>575 | <ul> <li>Guidance on accessing the CGM trace, either through a manufacturer-provided software<br/>app or via a study-provided CGM receiver unit, or via a personal insulin pump if<br/>participants use a pump that integrates with the study CGM</li> </ul> |
| 576<br>577 | • Parents will be asked to perform fingerstick blood glucose measurements in accordance with the labeling of the study CGM device |

A copy of the study CGM user's guide will be provided to the participant's parents.

578

546

547

3.1 CGM Run-in Phase Overview

## 579 **3.3 Blood Glucose and Ketone Testing**

- Participants will receive supplies for blood glucose and ketone testing.
- Blood glucose testing

582

583

584

585

586

587

590

592

593

594

595

596

597

- Participants will be provided with a study blood glucose meter, test strips, and standard control solution to perform quality control (QC) testing at home per manufacturer guidelines.
  - o All study blood glucose meters will be QC tested with control solution if available prior to dispensation and during all office visits. A tested meter will not be used in a study if it does not read within the target range at each concentration per manufacturer labeling.
- 588 o Participants will be reminded to use the study blood glucose meter for all fingerstick BGs during the study.
  - o Participants will be given guidelines for treatment of low or high blood glucose.
- Blood ketone testing
  - o Participants will be provided with a study blood ketone meter, test strips, standard control solution to perform QC testing at home per manufacturer guidelines, and software/hardware needed to download meter datafiles.
  - All study blood ketone meters will be QC tested with control solution if available prior to dispensation and during all office visits. A tested meter will not be used in a study if it does not read within the target range at each concentration per manufacturer labeling.
- 598 Participants will be instructed to perform blood ketone testing as described in section 7.1.6.
- o Participants will be given guidelines for treatment of elevated blood ketones
- Participants will be required to have glucagon at home. Participants who currently do not have one will be given a prescription for glucagon (either emergency kit or nasal glucagon per investigator discretion for participants over 4 years of age).

## 3.4 Assessment of Successful Completion of the Run-in Phase

- 604 Enrolled participants will have a follow-up visit or videoconference approximately 14 days after
- initiation of the run-in phase to assess progress or successful completion of the phase. If needed,
- one or more interim visits or videoconference/phone contacts may occur to assist the participant
- with any CGM use issues. Procedures will include downloading of the study CGM data and the
- 608 following:
- Assessment of compliance with the use of CGM for at least 11 out of the prior 14 days
- Assessment of skin reaction in areas where a CGM sensor was worn or other safety issues
- associated with CGM use
- Assessment of eligibility to continue to the randomized control trial (RCT) phase of the study

## 614 Participants Using a Personal CGM at Enrollment

- Participants who had currently been using a personal CGM at the time of enrollment (but did not
- meet requirements to skip run-in) and satisfy the CGM use criteria above without any major safety
- 617 issues and otherwise meet study eligibility requirements can be randomized.
- Participants who fail to meet the minimum CGM use requirement, or who the investigator believes
- may benefit from an extension of the CGM run-in period, may at the investigator's discretion be
- allowed to continue CGM run-in for a maximum of two additional 2-week periods. These
- participants will have a follow-up visit or videoconference approximately 14 days after each prior
- assessment for a reassessment using the same procedures as described above.
- Participants who do not meet CGM use requirements after three 2-week periods of CGM run-in or
- otherwise fail to meet study eligibility requirements will be withdrawn from the study.
- 625 Participants Not Using a Personal CGM at Enrollment
- Participants who had not currently been using a personal CGM at the time of enrollment will be
- assessed as described above. If there are no major safety issues and the investigator believes that
- 628 the participant will remain adherent to use of the study CGM, the participant will be asked to
- 629 continue the run-in phase for an additional 2-week period to establish baseline glycemic control
- while using the study CGM. These participants will have a follow-up visit or videoconference
- approximately 14 days for a second follow-up visit with the same visit procedures as described
- 632 above.
- Participants who fail to meet the minimum CGM use requirement at the second follow-up, or who
- the investigator believes may benefit from a further extension of the CGM run-in period, may at
- the investigator's discretion be allowed to continue CGM run-in for one additional 2-week period.
- These participants will have a follow-up visit or videoconference approximately 14 days after the
- second follow-up visit for a reassessment using the same procedures as described above.
- Participants who do not meet CGM use requirements after three 2-week periods of CGM run-in or
- otherwise fail to meet study eligibility requirements will be withdrawn from the study.

## 640 **3.5 Optimization of Insulin Therapy**

- Data will be obtained from CGM and/or pump downloads prior to CGM run-in review contacts.
- Adjustments to pump settings (basal rates, correction factor, insulin-to-carbohydrate ratio, etc.) or
- 643 injection strategies will be made in response to major trends observed in the CGM data, with
- 644 flexibility for clinicians to adhere to guidelines and practices established at each individual practice
- rather than a fixed set of heuristics for all clinical centers.

# **Chapter 4: Randomization Visit**

| 647 | 4.1 Visit Timing |
|---|---|
| 648<br>649<br>650<br>651 | The visit, which may be in-clinic or virtual, may occur on the same day as the Screening or Run-<br>in Review Visit, or on a subsequent day. If deferred, the randomization visit should occur no more<br>than 14 days after successful completion of the run-in phase or within 14 days of screening if run-<br>in is skipped. |
| 652 | 4.1.1 Randomization |
| 653 | Eligible participants will be randomly assigned to one of two treatment groups in a 2:1 ratio: |
| 654 | 1. Control-IQ Closed-Loop Control (CLC) Group |
| 655 | 2. Standard Care (SC) Group |
| 656<br>657<br>658 | The participant's randomization group assignment is determined by completing a Randomization Visit case report form on the study website. The randomization list will use a permuted block design, stratified by clinical center. |
| 659<br>660<br>661<br>662 | The participant will be included in the data analysis regardless of whether or not the protocol for the assigned randomization group is followed. Thus, the investigator must not randomize a participant until he/she is convinced that the participant/parent will accept assignment to either of the two groups. |
| 663<br>664<br>665 | It was decided that it was more important to stratify randomization by clinical center than by factors such as baseline time in range, HbA1c, or device use since these factors will be easier to adjust for in analysis than will clinical center. |
| 666 | 4.1.2 Baseline HbA1c Determination |
| 667<br>668<br>669 | A capillary blood sample will be obtained for baseline HbA1c determination. Capillary collection supplies will be provided to the participant within 3 days of randomization. This may occur either in-person at the clinic, or via delivery by other means (personal delivery, overnight shipment, etc.). |

## **Chapter 5: Main Study Procedures**

#### 671 5.1 Visit and Contact Schedule

670

673

676

677

679

688

672 During the RCT period, visits and contacts will be scheduled as outlined in Table 3 below:

## **Table 3: RCT Visit and Phone Contact Schedule**

| Target Day/Week | Contact Type <sup>1</sup> | Target/Allowable Window (around Target Day/Week) |
|---|---|---|
| 3 days <sup>2</sup> | VC/P | ± 2 days |
| 1 week | P | ± 2 days |
| 2 weeks | VC/V | ± 4 days |
| 6 weeks | VC/V | ±7 days |
| 10 weeks | P | ±7 days |
| 13 weeks | VC/V | ±7 days |

674 <sup>1</sup> Contact Types are defined as Clinic Visit (V), Videoconference (VC), or Phone call (P); Phone calls may be replaced by 675

Videoconferences or Clinic Visits and Videoconferences may be replaced by Clinic Visits at investigator discretion

<sup>2</sup> Only for participants on MDI at enrollment assigned to the CLC group; timing will be with respect to the start of home use of the study system, rather than with respect to the start of the RCT

678 Additional contacts or visits may occur as needed.

## 5.2 CGM Initiation and Training

- 680 Participants who skipped CGM run-in will be provided with study CGM supplies and training as
- 681 described in section 3.2 and instructed to use the study CGM on a daily basis. Participants
- 682 currently using a personal CGM identical to the study CGM may skip the training.
- 683 Provision of CGM supplies and training should be completed within 3 days of randomization.

#### 684 5.3 Procedures for the CLC Group

- 685 The study pump, associated supplies, and training will be provided to participants assigned to the
- 686 CLC group within 3 days of randomization. Dispensation of supplies may occur either in-person
- 687 at the clinic, or via delivery by other means (personal delivery, overnight shipment, etc.).

## 5.3.1 Study Pump Training

- 689 Parents of participants will receive study pump training by a qualified trainer. The participating
- 690 child will participate in training sessions to the degree judged appropriate by the parent and
- 691 trainer. Pump training (in-person or via videoconference) will be provided by a qualified trainer
- 692 to all CLC Group participants.
- 693 Parents will be fully instructed on the study insulin pump. The trainer will discuss differences from
- 694 the participant's personal pump, if applicable, in important aspects such as calculation of insulin
- 695 on board and correction boluses and optional additional topics such as: infusion site initiation,

- cartridge/priming procedures, setting up the pump, charging the pump, navigation through menus,
- bolus procedures including stopping a bolus, etc.
- Parents will be instructed to change the study insulin pump infusion set at least once every 3 days
- or per manufacturer guidelines, whichever is shorter.
- Parents will be trained to use the bolus calculator following the standard t:slim X2 training if they are not already using the t:slim X2 bolus calculator. Parent/guardians with prior
- education/experience with using this bolus calculator will be offered refresher training.
- The study team will assist the parent in study pump infusion site initiation and will start the participant on the study pump. The study pump will be programmed with the participant's usual basal rates and pump parameters, if applicable. The participant's personal pump, if any, will be removed.
  - The parent will be supervised with the study pump during at least one meal or snack bolus to ensure participant understanding of the pump features.
    - The parent will be encouraged to review the literature provided with the pump and infusion sets after the training is completed.
  - The parent will be trained on severe hypoglycemia emergency procedures including removal of the study pump and administration of glucagon.
- 713 Pump training specific to the Control-IQ Technology functions will include:
- How to turn on and off Control-IQ technology.
- How to understand when Control-IQ is increasing or decreasing basal rates.
- How to administer a meal or correction boluses
- What to do when exercising while using the system
- How to enable the sleep function and set the sleep schedule
- The parent will be assessed for understanding of the system interface and how to react to safety/alert messages.
- 721 The parent will be given a User Guide as a reference.

## 722 5.3.2 Initiation of Pump by MDI Participants

- 723 For MDI participants being started on the study pump, an initial basal insulin profile will be
- customized on a per-participant basis. Total daily insulin dose will be reduced by approximately
- 725 20% as a general rule, with a recommended method outlined in a separate procedures' manual.
- 726 Further adjustments to total daily dose (TDD) and intraday basal rate profile may be made during
- 727 the initial 2-week use period.

707

708

709

710

711

- Participants and parent(s) will complete training on the study pump as described above, with
- additional emphasis on topics relevant to new pump users, such as infusion site initiation,
- cartridge/priming procedures, setting up the pump, charging the pump, navigation
- through menus, bolus procedures including stopping a bolus, etc.
- The study team will assist the participant/parent in study pump infusion site initiation and will start
- the participant on the study pump. The study pump will be programmed with the participant's
- 734 insulin requirements.

# 735 **5.3.3 System Use Guidelines**

- 736 The participant/parent will be instructed to use the system in closed-loop mode except if insulin is
- delivered by any means other than the study pump (e.g. injection of subcutaneous insulin via
- 738 syringe in the event of infusion site failure). If insulin is delivered by any means other than the
- study pump, the parent will be instructed to turn off Control-IQ for approximately four hours.
- The parent will also be instructed to contact study staff if the participating child has illness with
- an elevated temperature >101.5 degrees Fahrenheit (38.6 degrees Celsius), other periods of
- significant illness, or during periods of use of medications such as epinephrine for the emergency
- 743 treatment of a severe allergic reaction or asthma attack in addition to use of oral or injectable
- glucocorticoids to determine if closed-loop use should be temporarily discontinued.
- Parents will be provided with sufficient supplies to last until the subsequent visit.
- Parents will be provided with contact information and will be asked to call the study clinical staff
- for any health-related issues and for technical issues with the system. Participants may use the
- 748 study pump without Control-IQ activated and study CGM during periods of component
- 749 disconnections or technical difficulties. Parents will also receive study staff contact information
- 750 to ask any questions they may have during the study.
- 751 Study staff will discuss with the parent that routine contact is required and will make arrangements
- with the parent for the contacts. If the parent cannot be reached, the participant's other contact
- methods will be utilized, including the emergency contact. Parents who are not compliant with
- 754 the arranged contacts on two separate occasions may be discontinued at the discretion of the
- 755 investigator.

762

- Upon completion of the CGM or study pump training components, as applicable, study staff will
- document, using a checklist, that the parent is familiar with the functions/features/tasks addressed
- 758 during the training.
- Parents will be provided Hypoglycemia, Hyperglycemia and Ketone Guidelines (section 8.2) for
- 760 when their glucose levels are >300 mg/dL for more than 90 minutes or >400 mg/dL at any time or
- 761 <70 mg/dL or ketones  $\ge$ 1.0 mmol/L.

## 5.3.4 Home Use of the Study System

- After training on the study system has been completed, participants will proceed with home use
- 764 (meaning free-living use at school, home, etc.) of the study pump.
- Parents may use available manufacturer-provided software and features of the study CGM related
- to mobile data access or remote monitoring, but will be instructed not to use any third-party
- 767 components for this purpose.

#### 768 5.3.5 Study Device Download

- Parents will be instructed to download the study CGM and pump and ketone meter prior to each
- phone or videoconference contact or on at least an every 4-week basis throughout the remainder
- of the study.

#### **5.3.6 3-Day Phone Contact**

- For participants who were on MDI at the time of enrollment, study staff will perform a phone call
- or videoconference with the parent within 3 ( $\pm 2$ ) days following initiation of study pump use.
- 775 The following will occur:
- Assessment of compliance with study device use by review of any available device data
- Assessment of adverse events, adverse device effects, and device issues
- Study staff will answer any questions related to device use and follow the procedure for insulin pump optimization described above using the study CGM available data from the previous two weeks.

### **5.3.7 1-Week Phone Contact**

- Study staff will perform a phone call/videoconference with the parent within 7 ( $\pm 2$ ) days following
- 783 randomization.

785

- 784 The following will occur:
  - Assessment of compliance with study device use by review of any available device data
- Assessment of adverse events, adverse device effects, and device issues
- Study staff will answer any questions related to device use and follow the procedure for insulin pump optimization described above using the study CGM available data from the previous two weeks.

#### 790 **5.3.8 2-Week Visit**

- Participants will have a follow-up visit 14 ( $\pm$ 4) days from the date of randomization.
- The parent will be offered review training to address any questions on the use of the study device
- 793 including meal bolus strategies and strategies related to pump use and exercise.
- 794 The following will occur:
- Assessment of compliance with study device use by review of any available device data
- Assessment of adverse events, adverse device effects, and device issues
- Study staff will answer any questions related to device use and follow the procedure for insulin pump optimization described above using the study CGM available data from the previous two weeks.

• At in-clinic visits, the blood glucose meter and study ketone meter will be downloaded and QC tested with control solution.

# **5.4 Procedures for the SC Group**

- Participants in the SC group will continue to use their existing insulin therapy (personal pump or
- MDI) for the treatment of their diabetes, in conjunction with use of the study CGM, study blood
- glucose meter, and study ketone meter.
- 806 If a participant is using a pump with an LGS/PLGS feature, he/she will be allowed to continue
- 807 using this feature during the trial.
- Parents may use available manufacturer-provided software and features of the study CGM related
- 809 to mobile data access or remote monitoring, but will be instructed not to use any third-party
- 810 components for this purpose.

### 811 **5.4.1 Study Device Data Download**

- Parents will be instructed to upload/email data from the study CGM and study ketone meter using
- 813 commercially available software prior to each phone or videoconference contact below for
- 814 clinician review. Parents will be provided with any software and hardware needed to perform
- 815 these data uploads.

#### 816 **5.4.2 1-Week Phone Contact**

- Study staff will perform a phone call/videoconference with the participant  $7(\pm 2)$  days following
- 818 randomization.
- 819 The following will occur:
- Assessment of compliance with study device use by review of any available device data
- Assessment of adverse events, adverse device effects, and device issues
- Study staff will answer any questions related to device use

#### 823 **5.4.3 2-Week Visit**

- Participants will have a follow-up visit 14 ( $\pm$ 4) days from the date of randomization.
- The parent will be offered review training on the use of SC during the remainder of the study,
- including meal bolus strategies and strategies related to exercise.
- 827 The following will occur:

- Assessment of compliance with study device use by review of any available device data
- Assessment of adverse events, adverse device effects, and device issues
- Study staff will review uploaded CGM data, answer any questions related to device use, and provide any recommendations for insulin therapy adjustment.

- If visit is in-clinic, the study blood glucose meter and study ketone meter will be downloaded and QC tested.
- The parent will be instructed to upload data from the study CGM and ketone meter at least once
- every 4 weeks for the remainder of the study.

#### 5.5 Follow-up Visits and Phone Contacts for Both Groups

- After the first 2 weeks, the schedule for remaining follow-up contacts is the same for both
- treatment groups. Study staff will discuss with the parent that periodic contact is required and will
- 839 make arrangements with the parent for the contacts. If the parent cannot be reached, the
- participant's other contact methods will be utilized, including the emergency contact.

#### 841 **5.5.1 Visits**

- A follow-up in-clinic visit will occur at 6 weeks ( $\pm 7$  days). The following procedures are
- performed in both groups, unless otherwise specified below:
- Assessment of compliance with study device use by review of any available device data
- Assessment of adverse events, adverse device effects, and device issues
- Download of device data (study system or personal pump and study CGM, study BG meter, study
- ketone meter); in the case of videoconferences, participants will upload or email available data
- prior to the visit, including CGM, pump, and ketone meter, so that clinic staff can review and
- 849 download the data

854

855

856

858

#### **5.5.2 Phone Contacts**

- A follow-up phone call or videoconference will occur at 10 weeks ( $\pm 7$  days). At the discretion of
- the investigator, this scheduled phone contact may be replaced by an in-clinic visit.
- The following procedures are performed in both treatment groups:
  - Review of available CGM, ketone meter, and/or system data to identify any safety issues associated with current insulin therapy and diabetes management approach
  - Assessment of adverse events, adverse device effects, and device issues
- Additional phone contacts may be performed as needed.

#### 5.5.3 Optimization of Insulin Therapy

- 859 If needed for safety reasons at the criteria of the physician at each clinical center, optimization may
- be done via phone contacts, videoconferences, or in-clinic visits.
- Data will be obtained from CGM and/or pump downloads during the contact. Adjustments to pump
- settings (basal rates, correction factor, insulin-to-carbohydrate ratio, etc.) or injection strategies
- will be made in response to major trends observed in the CGM data, with flexibility for clinicians
- to adhere to guidelines and practices established at each individual practice rather than a fixed set
- of heuristics for all clinical centers.

#### 866 **5.5.4 13-Week Visit**

- All participants will have a 13-Week (±7 days) visit during which the following will occur:
- Collection of a blood sample to send to the central laboratory for HbA1c determination.
- Completion of questionnaires
- Weight and height measurements will be repeated
- Assessment of adverse events, adverse device effects, and device issues
- Download of device data (study system or personal pump and study CGM, study BG meter, study ketone meter) as available

# **5.6 Early Termination Visit (If Applicable)**

- Participants will be asked to come for an end of study visit in the event of withdrawal or early
- 876 termination.

880

#### 877 **5.7** Unscheduled Visits

- Participants may have unscheduled visits during the study period if required for additional device
- training or other unanticipated needs per the study investigator discretion.

# **Chapter 6: Extension Phase Procedures**

- 882 At the conclusion of the 13-week RCT, all participants will use the Control-IQ closed-loop 883 system during a 13-week Extension Phase.
- 884 An updated version of the Control-IQ system with enhanced usability will be used during the
- 885 Extension Phase. Participants assigned to the SC group during the RCT period will receive
- 886 training based on the updated pump as described below. Participants assigned to the CLC group
- 887 will receive a brief training session to review any new or changed features of the pump.
- Initiation of the updated Control-IQ pump may be deferred by up to 2 weeks if needed, with the 888
- 889 participant continuing on the treatment used during the RCT period during this time and the
- 890 overall duration of the Extension Phase increasing by up to 2 weeks.

#### 6.1 Visit and Contact Schedule

881

891

892

893

894

895

896

897 898

899

900

During the Extension period, visits and contacts will be scheduled as outlined in Table 4 below:

#### Table 4: Extension Phase Visit and Phone Contact Schedule

| Target Day/Week <sup>1</sup> | Contact Type <sup>2</sup> | Target/Allowable Window (around Target Day/Week) |
|---|---|---|
| 13 weeks + 3 days | VC/P | ± 2 days |
| 14 weeks | P | ± 2 days |
| 15 weeks | VC/V | ± 4 days |
| 19 weeks | VC/V | ±7 days |
| 23 weeks | P | ±7 days |
| 26 weeks | VC/V | ±7 days |

<sup>&</sup>lt;sup>1</sup> The "13 weeks" and subsequent visit targets reflect a participant who had no delay between the 13-week visit of the RCT and initiation of use of the updated Control-IO pump. Targets and associated windows may be shifted by up to 2 weeks for participants whose initiation is delayed.

<sup>2</sup> Contact Types are defined as Clinic Visit (V), Videoconference (VC), or Phone call (P); Phone calls may be replaced by

#### **6.2 Study Pump Initiation**

- 901 Participants assigned to the SC group during the initial 13-Week RCT period will initiate use of
- 902 the updated study pump either the same day as the 13-Week visit or within 2 weeks of this visit.
- 903 The procedures described in section 5.3 above will be followed to initiate these participants on
- 904 the study pump.
- 905 Participants assigned to the CLC group during the RCT period will switch to the updated version
- 906 of the Control-IQ system and will receive training on its new features. This will occur either the
- 907 same day as the 13-Week visit or within 2 weeks of this visit.

Videoconferences or Clinic Visits and Videoconferences may be replaced by Clinic Visits at investigator discretion

# 908 6.3 Visits, Videoconferences, and Phone Calls for All Participants

# 909 **6.3.1 13-Week + 3-Day Phone Contact**

- Study staff will perform a phone call or videoconference with the parent within 3 ( $\pm 2$ ) days
- 911 following initiation of Extension Phase study pump use. Procedures will mirror those described in
- 912 section 5.3.6 above.

#### 913 **6.3.2 14-Week Phone Contact**

- Participants will have a phone call or videoconference at 14 Weeks (±2 days). Procedures will
- 915 mirror those described in section 5.3.7 above.

#### 916 **6.3.3 15-Week Visit**

- Participants will have a follow-up visit at 15 Weeks (±4 days). Procedures will mirror those
- 918 described in section 5.3.8 above.

#### 919 **6.3.4 19-Week Visit**

- A follow-up in-clinic visit will occur at 19 weeks ( $\pm 7$  days). Procedures will mirror those
- 921 described in section 5.5.1 above.

#### 922 **6.3.5 23-Week Phone Call**

- A follow-up phone call will occur at 23 weeks ( $\pm 7$  days). Procedures will mirror those described
- 924 in section 5.5.2 above.

#### 925 **6.3.6 26-Week Visit**

- A follow-up in-clinic visit will occur at 26 weeks ( $\pm 7$  days). Procedures will mirror those
- 927 described in section 5.5.4 above.
- Participants will have the opportunity to participate in Focus Group sessions as described in
- 929 section 9.3 below.
- Participants will be given the option to continue use of the Control-IQ closed-loop system during
- an additional Extended Use period as described in the next chapter. Participants who do not wish
- 932 to continue to the Extended Use period will be switched back to the insulin pump or MDI
- 933 therapy that was in use prior to the study.

## 934 **6.3.7 Optimization of Insulin Therapy**

- 935 If needed for safety reasons at the criteria of the physician at each clinical center, optimization
- may be done via phone contacts, videoconferences, or in-clinic visits as described in section
- 937 5.5.3 above.

#### 938 **6.4 Unscheduled Visits**

- Participants may have unscheduled visits during the study period if required for additional device
- training or other unanticipated needs per the study investigator discretion.

# 6.5 Participant Access to Study Device at Study Closure

Participants not continuing to the Extended Use period will return all investigational study devices and supplies (insulin pump, CGM and related supplies). Participants may keep the study ketone meter and study glucometer if these devices are not marked for investigational use only.

945

# **Chapter 7: Extended Use Period Procedures**

- At the 26-Week Visit of the Extension Phase, participants will be given the option to continue use of the Control-IQ closed-loop system during an additional Extended Use period. Participants who completed the 26-Week Visit before the addition of this Extended Use period to the study
- protocol will be eligible to rejoin the study and participate as long as they completed their 26-
- Week Visit within the prior 4 months.
- The same version of the Control-IQ system in use during the 13-Week Extension Phase will be
- 953 used during the Extended Use period.
- 954 Informed Consent will be obtained from eligible participants who are interested in participating
- in the Extended Use period. The informed consent process will mirror the process described
- 956 above in section 2.1.1.

#### 7.1 Visit and Contact Schedule

- During the Extended Use period, visits and contacts will be scheduled as outlined in Table 5
- 959 below:

957

960

965

967

946

**Table 5: Extended Use Period Visit and Phone Contact Schedule** 

| Target Day/Week with<br>respect to initiation of<br>Extended Use period | Contact Type <sup>1</sup> | Target/Allowable Window<br>(around Target Day/Week) |
|---|---|---|
| 0 days (Retraining) <sup>2</sup> | VC/V | N/A |
| 3 days <sup>2</sup> | VC/P | ± 2 days |
| 1 week <sup>2</sup> | VC/P | ± 2 days |
| 13 weeks | VC/V | ±7 days |
| 26 weeks | VC/V | ±7 days |
| Final Visit | VC/V | N/A |

<sup>961</sup> Contact Types are defined as Clinic Visit (V), Videoconference (VC), or Phone call (P); Phone calls may be replaced by

# 7.2 Visits, Videoconferences, and Phone Calls for Participants Re-Initiating Study Pump

# 966 Use After a Gap in Use

#### 7.2.1 Study Pump Retraining Visit

- Participants who had a gap between the 26-Week Visit and the initiation of the Extended Use
- 969 period during which they reverted to MDI or personal pump insulin therapy will have a visit to
- 970 receive retraining on the study pump prior to re-initiation of study pump use.

Videoconferences or Clinic Visits and Videoconferences may be replaced by Clinic Visits at investigator discretion

 <sup>2</sup> Only for participants who had a gap between the 26-Week Visit and the initiation of the Extended Use period during which they stopped use of the study pump and reverted to MDI or personal pump insulin therapy

- The procedures described in section 5.3 above will be followed to re-initiate these participants on
- 972 the study pump.
- **7.2.2 3-Day Phone Contact**
- 974 Study staff will perform a phone call or videoconference with the parent within 3 (±2) days
- 975 following re-initiation of study pump use. Procedures will mirror those described in section 5.3.6
- 976 above.
- **7.2.3 1-Week Phone Contact**
- Participants will have a phone call or videoconference within 7 days (±2 days) following re-
- 979 initiation of study pump use. Procedures will mirror those described in section 5.3.7 above.
- 980 7.3 Visits, Videoconferences, and Phone Calls for All Participants
- 7.3.1 13-Week Visit and Subsequent Visits Every 13 Weeks
- A follow-up in-clinic visit will occur 13 weeks ( $\pm 7$  days) after the start of the Extended Use period.
- The following procedures will be performed in both groups:
- Collection of a blood sample to send to the central laboratory for HbA1c determination
- Assessment of compliance with study device use by review of any available device data
- Assessment of adverse events, adverse device effects, and device issues
- Download of device data (study system or personal pump and study CGM, study BG meter, study ketone meter); in the case of videoconferences, participants will upload or email available data prior to the visit, including CGM, pump, and ketone meter, so that clinic staff can review and download the data
- 991 Every 13 weeks (±7 days) thereafter, another follow-up clinic visit will occur involving the same
- procedures described above.
- 993 **7.3.2** Final Visit
- A final follow-up in-clinic or videoconference visit will occur no later than July 31, 2022.
- Procedures will mirror those described in section 7.3.1 above, except that no blood sample will
- 996 be collected.
- Participants will be switched back to the insulin pump or MDI therapy that was in use prior to
- 998 the study.
- 999 7.3.3 Optimization of Insulin Therapy
- 1000 If needed for safety reasons at the criteria of the physician at each clinical center, optimization
- may be done via phone contacts, videoconferences, or in-clinic visits as described in section
- 1002 5.5.3 above.

# 7.4 Unscheduled Visits

- Participants may have unscheduled visits during the study period if required for additional device
- training or other unanticipated needs per the study investigator discretion.
- 1006 7.5 Participant Access to Study Device at Study Closure
- 1007 Participant will return all investigational study devices and supplies (insulin pump, CGM and
- 1008 related supplies) at study closure. Participant may keep the study ketone meter and study
- glucometer if these devices are not marked for investigational use only.

#### **Chapter 8: Study Devices** 1010 1011 8.1 Description of the Investigational Device 1012 8.1.1 Insulin Pump 1013 The study system will include the Tandem t:slim X2 with Control-IQ technology. 1014 **8.1.2** Continuous Glucose Monitoring 1015 The study CGM will include Dexcom G6 transmitter and sensors. The CGM sensor will be 1016 replaced at least once every 10 days. 1017 **8.1.3 Blood Glucose Meter and Strips** 1018 Blood glucose levels will be measured using the study's blood glucose meter (glucometer) and the 1019 CGM device will be calibrated if needed using the study glucometer and strips in accordance with 1020 the manufacturer's labeling. 1021 8.1.4 Ketone Meter and Strips 1022 Blood ketone levels will be measured using the Abbott Precision Xtra meter and strips in 1023 accordance with the manufacturer's labeling. The blood glucose meter component of the Precision Xtra device will not be used. 1024 1025 8.1.5 Study Device Accountability Procedures 1026 Device accountability procedures will be detailed in the clinical center procedures manual. 1027 **8.1.6 Blood Ketone Testing** 1028 Participants to perform QC testing at home per manufacturer guidelines. 1029 All study blood ketone meters will be QC tested with control solution if available during all office 1030 visits. A tested meter will not be used in a study if it does not read within the target range at each concentration per manufacturer labeling. The participant will be instructed to contact study staff 1031 1032 for a replacement of the meter, test strips, and control solution if a meter fails QC testing at home. 1033 Participants will be instructed on how to perform blood ketone testing. 1034 Participants will be given guidelines for treatment of elevated blood ketones. 1035 8.2 Safety Measures 1036 8.2.1 CGM Calibration 1037 Throughout the study, participants will be instructed to calibrate the study CGM in accordance 1038 with manufacturer labelling.

# **8.2.2 System Failure**

- 1040 If the CGM signal becomes unavailable for more than 20 minutes consecutively, Control-IQ or
- 1041 closed loop will not operate to automatically adjust insulin. If the CGM is not connected, the
- system will revert to usual function of the pump and deliver insulin with the insulin dosing
- parameters programmed in the system for that individual. Resumption of Closed-Loop will
- occur automatically once CGM signal is available again.
- 1045 If the study system is unable to activate Control-IQ for any reason, the pump will automatically
- revert to preprogrammed basal insulin delivery without any need for instruction from the user.
- 1047 If the pump detects a system error that does not allow it to operate, the Malfunction Alarm will
- display and the participant will be instructed to contact Tandem Technical Support via the study
- 1049 team.

1061

# 1050 8.2.3 Hypoglycemia Threshold Alert and Safety Protocol

- During the course of the study, participants will be permitted to change the CGM low glucose
- threshold alert setting on their device or mobile app, but will be instructed to choose a value no
- less than 70 mg/dL.
- The t:slim X2 with Control-IQ system will issue a predictive hypoglycemia alert (Control-IQ Low
- Alert) when the system predicts BG <70 mg/dL within the next 15 minutes (<80 mg/dL when
- 1056 exercise mode is activated).
- 1057 If the participant receives a Control-IQ Low Alert, a message appears on the user interface (UI)
- that is accompanied by vibration followed by vibrations and/or sound if not acknowledged by the
- user in 5 minutes. This alert remains on the screen until acknowledged by the user. The user is
- prompted to test blood sugar and treat with carbs.

#### 8.2.4 Hyperglycemia Threshold Alert and Safety Protocol

- During the course of the study, participants will be permitted to change the CGM high glucose
- threshold alert setting on their device or mobile app, but will be instructed to choose a value no
- greater than 300 mg/dL.
- The t:slim X2 with Control-IO system will issue a predictive hyperglycemia alert (Control-IO
- High Alert) when the system has increased insulin delivery, but detects a CGM value above 200
- 1067 mg/dL and does not predict the value will decrease in the next 30 minutes.
- 1068 If the participant receives a Control-IQ High Alert, a message appears on the UI that is
- accompanied by vibration followed by vibrations and/or sound if not acknowledged by the user in
- 5 minutes. This alert remains on the screen until acknowledged by the user. The user is prompted
- to check the site for occlusion and test blood glucose.
- 1072 If a participant's CGM reading is >300 mg/dL for over 90 minutes or ≥400 mg/dL at any point, or
- if CGM reading is >250 mg/dL more than 3 hours after a meal, the participant took correction

- 1074 insulin, and CGM didn't decrease by at least 50 mg/dL, the participant will be instructed to take
- the following steps:
- 1076 Inspect infusion site for problems
- 1077 Perform a blood glucose meter check.
- 1078 If the blood glucose is >300 mg/dL, check for blood ketones with the study ketone meter.
- 1079 If the ketone level is ≥1.0 mmol/L, take correction insulin, change insulin (pump) infusion site and
- 1080 contact study staff.
- 1081 If a participant administers correction insulin via insulin syringe, participants will be instructed to
- turn Control-IQ off for approximately four hours.

# 1083 Chapter 9: Testing Procedures, Questionnaires, and Focus Groups

- 1084 **9.1 Laboratory Testing**
- 1085 **9.1.1 HbA1c:**
- Performed at the Randomization visit, 13-Week visit, and 26-Week visit
- Blood samples will be sent to the central laboratory for sample analysis using an NGSP approved
- 1088 method.
- 1089 **9.2 Ouestionnaires**
- The questionnaires listed below are completed by participants' parents at Screening, 13 weeks,
- and 26 weeks for all participants except as noted. The questionnaires will be family and age
- appropriate and are described briefly below. The procedures for administration are described in
- the clinical center procedures manual.
- 1094 Pediatric Quality of Life Parent
- 1095 Pediatric Inventory for Parents
- 1096 INSPIRE Survey Parent
- 1097 Pittsburgh Sleep Quality Index (PSQI) Parent
- 1098 Fear of Hypoglycemia Survey-Parents (HFS-P)
- 1099 Hypoglycemia Confidence Scale (HCS)
- 1100 System Usability Scale (SUS) (Closed-Loop participants only at 13 and 26 weeks)
- 1101 Administration time is approximately 35 minutes.
- 1102 9.2.1 PedsQL Diabetes Module Parent
- This is a 32-item scale developed and validated for the measurement of diabetes-specific quality
- of life. Participants record the extent to which their child experienced each of 32 problems
- related to diabetes in the prior month.
- 1106 Administration time is approximately 5 minutes.
- 1107 9.2.2 Pediatric Inventory for Parents
- This is a widely-used, 42-item measure of parenting stress designed for parents of youth with
- type 1 diabetes.
- 1110 Administration time is approximately 6 minutes.
- 1111 9.2.3 INSPIRE Survey Parent
- The INSPIRE (<u>Insulin Delivery Systems</u>: <u>Perceptions</u>, <u>Ideas</u>, <u>Reflections and Expectations</u>) survey
- was developed to assess various aspects of a user's experience regarding automated insulin

- delivery for both patients and family members. The surveys include various topics important to
- patients with type 1 diabetes and their family members based upon >200 hours of qualitative
- interviews and focus groups. The parent pre-assessment survey and parent post-assessment survey
- both contain 19 items. Response options for all surveys include a 5-point Likert scale from strongly
- agree to strongly disagree, along with an N/A option.
- 1119 Administration time is approximately 5 minutes.
- 9.2.4 Pittsburgh Sleep Quality Index (PSQI) Parent
- An abbreviated 9-question version of the Pittsburgh Sleep Quality Index (PSQI), a validated tool
- for assessing self-reported sleep quantity and quality, will be completed by parents. Seven
- component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The
- 1124 component scores are summed to produce a global score (range 0 to 21). Higher scores indicate
- worse sleep quality.
- Administration time is approximately 3 minutes.
- 1127 9.2.5 Hypoglycemia Fear Survey-Parent (HFS-P)
- The Hypoglycemia Fear Survey-Parent is a validated tool of 25 items to assess parents' anxiety
- and behavior concerning possible hypoglycemia. Items are rated on a 5-point Likert scale
- 1130 (0=never, 4=always), with higher scores indicating higher fear of hypoglycemia.
- 1131 Administration time is approximately 4 minutes.
- 1132 9.2.6 Hypoglycemia Confidence Scale
- The scale comprises 8 items and measures confidence hypoglycemia can be treated or prevented
- in various situations.
- Administration time is approximately 3 minutes.
- 1136 9.2.7 System Usability Scale (SUS)
- 1137 The System Usability Scale (SUS) is a 10-item questionnaire that measures the overall usability
- of a system. It is a valid and reliable measure of the perceived usability of a system and is
- technology-agnostic. The questionnaire presents statements with five response options (anchoring
- the options from strongly disagree to strongly agree) and asks users to rate their agreement to the
- statements. User scores are transformed into a composite score, from 0 to 100, and this score is
- taken as an overall measure of the system's usability; higher scores indicate better perceived
- 1143 usability.
- 1144 Administration time is approximately 5 minutes.
- 1145

#### 9.3 Focus Groups

- Focus groups will be completed following the 26-Week Visit. The focus groups will be conducted
- virtually using HIPAA-approved software.
- Focus groups will include 3-5 individuals and a script of open-ended questions to gather feedback
- and reactions to the closed loop system, the clinical trial, and QoL changes. There will also be time
- for discussion of content raised by parents. If parents are able to have the child participant attend
- briefly to answer a few questions, this will be attempted.
- Sessions will be audio- and video-taped and transcribed by a professional transcription service.
- Otherwise, these recordings will not be shared for any non-study purposes. Transcriptions will use
- a code for participants, such as "Participant 1", and will not contain names or other identifiers of
- 1156 participants.

# 1157 Chapter 10: Unanticipated Problem, Adverse Event, and Device Issues

| 1158 | Reporting |
|---|---|
| 1159 | 10.1 Unanticipated Problems |
| 1160<br>1161<br>1162<br>1163<br>1164 | Site investigators will promptly report to the Coordinating Center on an eCRF all unanticipated problems meeting the criteria below. Problems meeting IRB reporting requirements will be reported to the IRB within 7 calendar days of the site becoming aware of the problem. For this protocol, an unanticipated problem is an incident, experience, or outcome that meets all of the following criteria: |
| 1165<br>1166<br>1167<br>1168 | • Unexpected (in terms of nature, severity, or frequency) given (a) the research procedures that are described in the protocol related documents, such as the IRB-approved research protocol and informed consent document; and (b) the characteristics of the subject population being studied |
| 1169<br>1170<br>1171 | • Related or possibly related to participation in the research (possibly related means there is a reasonable possibility that the incident, experience, or outcome may have been caused by the procedures involved in the research) |
| 1172<br>1173<br>1174 | <ul> <li>Suggests that the research places participants or others at a greater risk of harm than was<br/>previously known or recognized (including physical, psychological, economic, or social<br/>harm)</li> </ul> |
| 1175<br>1176<br>1177<br>1178<br>1179<br>1180<br>1181 | The Coordinating Center also will report to the IRB all unanticipated problems not directly involving a specific site such as unanticipated problems that occur at the Coordinating Center or at another participating entity such as a pharmacy or laboratory. These instances must be reported to the JCHR IRB within seven calendar days of recognition. The Director of the Human Research Protection Program will report to the appropriate regulatory authorities if the IRB determines that the event indeed meets the criteria of an Unanticipated Problem requiring additional reporting. |
| 1182 | 10.2 Adverse Events |
| 1183 | 10.2.1 Definitions |
| 1184<br>1185 | Adverse Event (AE): Any untoward medical occurrence in a study participant, irrespective of the relationship between the adverse event and the device(s) under investigation. |
| 1186 | Serious Adverse Event (SAE): Any untoward medical occurrence that: |
| 1187 | Results in death. |
| 1188<br>1189 | Is life-threatening; (a non-life-threatening event which, had it been more severe, might have become life-threatening, is not necessarily considered a serious adverse event). |
| 1190 | Requires inpatient hospitalization or prolongation of existing hospitalization. |

- Results in persistent or significant disability/incapacity or substantial disruption of the ability to
- 1192 conduct normal life functions (sight threatening).
- 1193 Is a congenital anomaly or birth defect.
- 1194 Is considered a significant medical event by the investigator based on medical judgment (e.g., may
- 1195 jeopardize the participant or may require medical/surgical intervention to prevent one of the
- outcomes listed above).
- 1197 <u>Unanticipated Adverse Device Effect (UADE):</u> Any serious adverse effect on health or safety or
- any life-threatening problem or death caused by, or associated with, a device, if that effect,
- problem, or death was not previously identified in nature, severity, or degree of incidence in the
- investigational plan or application (including a supplementary plan or application), or any other
- unanticipated serious problem associated with a device that relates to the rights, safety, or welfare
- 1202 of participants (21 CFR 812.3(s)).
- 1203 Adverse Device Effect (ADE): Any untoward medical occurrence in a study participant which the
- device may have caused or to which the device may have contributed (Note that an Adverse Event
- Form is to be completed in addition to a Device Deficiency or Issue Form, unless excluded from
- reporting as defined in section 10.3). An event that occurs solely due to participant (i.e., user)
- error in which the device functions properly generally will not be considered an ADE unless it is
- determined that the instructions on the screen of the device or user manual (or similar training
- materials) may have contributed to the event (note: the event may still meet criteria for reporting
- 1210 as an adverse event).
- 1211 <u>Device Complaints and Malfunctions:</u> A device complication or complaint is something that
- happens to a device or related to device performance, whereas an adverse event happens to a
- participant. A device complaint may occur independently from an AE, or along with an AE.
- 1214 An AE may occur without a device complaint or there may be an AE related to a device complaint.
- 1215 A device malfunction is any failure of a device to meet its performance specifications or otherwise
- perform as intended. Performance specifications include all claims made in the labeling for the
- device. The intended performance of a device refers to the intended use for which the device is
- labeled or marketed. (21 CFR 803.3). Note: for reporting purposes, sites will not be asked to
- distinguish between device complaints and malfunctions.

#### 1220 **10.2.2** Reportable Adverse Events

- 1221 For this protocol, a reportable adverse event includes any untoward medical occurrence that meets
- one of the following criteria:
- 1223 1. An SAE or an AE associated with a visit to a hospital emergency department
- 1224 2. An ADE as defined in section 10.2.1, unless excluded from reporting in section 10.3
- 1225 3. An AE as defined in section 10.2.1 occurring in association with a study procedure
- 4. An AE as defined in section 10.2.1 not related to a device issue which leads to temporary or permanent discontinuation of a study device
- 5. An AE as defined in section 10.2.1 that affects the participant's ability to complete any study procedures

- 1230 6. Hypoglycemia meeting the definition of severe hypoglycemia as defined below
- 7. Diabetic ketoacidosis (DKA) as defined below or in the absence of DKA, a hyperglycemic or
- ketosis event meeting the criteria defined below
- Hypoglycemia and hyperglycemia not meeting the criteria below will not be recorded as adverse
- events unless associated with an Adverse Device Effect. Skin reactions from sensor placement are
- only reportable if severe and/or required treatment.
- 1236 All reportable AEs—whether volunteered by the participant, discovered by study personnel during
- questioning, or detected through physical examination, laboratory test, or other means—will be
- reported on an AE form online. Each AE form is reviewed by the Medical Monitor to assess safety
- and to verify the coding and the reporting that is required.

# 1240 **10.2.3 Hypoglycemic Events**

- Hypoglycemia not associated with an Adverse Device Effect is only reportable as an adverse event
- when the following definition for severe hypoglycemia is met: the event required assistance of
- another person due to altered consciousness, and required another person to actively administer
- 1244 carbohydrate, glucagon, or other resuscitative actions. This means that the participant was
- impaired cognitively to the point that he/she was unable to treat himself/herself, was unable to
- verbalize his/ her needs, was incoherent, disoriented, and/or combative, or experienced seizure or
- loss of consciousness. These episodes may be associated with sufficient neuroglycopenia to
- induce seizure or loss of consciousness. If plasma glucose measurements are not available during
- such an event, neurological recovery attributable to the restoration of plasma glucose to normal is
- 1250 considered sufficient evidence that the event was induced by a low plasma glucose concentration.
- When a hypoglycemic event meets the above reporting requirements, a Hypoglycemia Form
- should be completed in addition to the Adverse Event Form. Severe hypoglycemia events should
- be considered to be serious adverse events with respect to reporting requirements.

#### 1254 **10.2.4** Hyperglycemic/Ketotic Events

- 1255 Hyperglycemia not associated with an Adverse Device Effect is only reportable as an adverse
- event when one of the following criteria is met:
- the event involved DKA, as defined by the Diabetes Control and Complications Trial (DCCT) and
- 1258 described below
- evaluation or treatment was obtained at a health care provider facility for an acute event involving
- 1260 hyperglycemia or ketosis, or the participant contacted the site and received guidance on how to
- manage the hyperglycemia/ketosis
- blood ketone level >1.0 mmol/L, even if there was no communication with a health care provider
- 1263 at the time of the event
- Hyperglycemic events are classified as DKA if the following are present:
- 1265 Symptoms such as polyuria, polydipsia, nausea, or vomiting;

- 1266 Serum ketones ≥1.5 mmol/L or large/moderate urine ketones;
- 1267 Either arterial blood pH <7.30 or venous pH <7.24 or serum bicarbonate (or CO<sub>2</sub>) <15; and
- 1268 Treatment provided in a health care facility
- 1269 When a hyperglycemia/ketotic qualifies as an SAE as defined in section 10.2.1, a
- 1270 Hyperglycemia/DKA Form should be completed in addition to the Adverse Event Form. Events
- meeting DKA criteria should be considered to be serious adverse events with respect to reporting
- requirements. Hyperglycemia events not meeting criteria for DKA generally will not be considered
- as serious adverse events unless one of the SAE criteria in section 10.2.1 is met.

# 1274 10.2.5 Relationship of Adverse Event to Study Device

- 1275 The study investigator will assess the relationship of any adverse event to be related or unrelated
- by determining if there is a reasonable possibility that the adverse event may have been caused by
- the study device.
- To ensure consistency of adverse event causality assessments, investigators should apply the
- following general guideline when determining whether an adverse event is related:
- 1280 Yes
- There is a plausible temporal relationship between the onset of the adverse event and the study
- intervention, and the adverse event cannot be readily explained by the participant's clinical state,
- intercurrent illness, or concomitant therapies; and/or the adverse event follows a known pattern of
- response to the study intervention; and/or the adverse event abates or resolves upon discontinuation
- of the study intervention or dose reduction and, if applicable, reappears upon re-challenge.
- 1286 <u>No</u>
- 1287 Evidence exists that the adverse event has an etiology other than the study intervention (e.g.,
- 1288 preexisting medical condition, underlying disease, intercurrent illness, or concomitant
- medication); and/or the adverse event has no plausible temporal relationship to study intervention.

#### 1290 **10.2.6** Severity (Intensity) of Adverse Events

- The severity (intensity) of an adverse event will be rated on a three point scale: (1) mild, (2)
- moderate, or (3) severe. A severity assessment is a clinical determination of the intensity of an
- event. Thus, a severe adverse event is not necessarily serious. For example, itching for several
- days may be rated as severe, but may not be clinically serious.
- MILD: Usually transient, requires no special treatment, and does not interfere with the participant's daily activities.
- MODERATE: Usually causes a low level of inconvenience, discomfort or concern to the participant and may interfere with daily activities, but is usually ameliorated by simple therapeutic measures and participant is able to continue in study.

- 1300 • SEVERE: Interrupts a participant's usual daily activities, causes severe discomfort, may 1301 cause discontinuation of study device, and generally requires systemic drug therapy or 1302 other treatment.
- 1303 10.2.7 Expectedness
- 1304 For a serious adverse event that is considered possibly related to study device, the Medical
- Monitor will classify the event as unexpected if the nature, severity, or frequency of the event is 1305
- not consistent with known risk information. 1306
- 1307 10.2.8 Coding of Adverse Events
- 1308 Adverse events will be coded using the MedDRA dictionary. To facilitate coding, the site will
- enter a preliminary MedDRA code which the Medical Monitor may accept or change (the Medical 1309
- 1310 Monitor's MedDRA coding will be used for all reporting). The Medical Monitor will review the
- 1311 investigator's assessment of causality and may agree or disagree. Both the investigator's and
- 1312 Medical Monitor's assessments will be recorded. The Medical Monitor will have the final say in
- determining the causality as well as whether an event is classified as a serious adverse event and/or 1313
- 1314 an unanticipated adverse device effect.
- 10.2.9 Outcome of Adverse Events 1315
- 1316 The outcome of each reportable adverse event will be classified by the investigator as follows:
- 1317 RECOVERED/RESOLVED – The participant recovered from the AE/SAE without sequelae.
- 1318 Record the AE/SAE stop date.
- 1319 RECOVERED/RESOLVED WITH SEQUELAE – The event persisted and had stabilized without
- change in the event anticipated. Record the AE/SAE stop date. 1320
- 1321 FATAL – A fatal outcome is defined as the SAE that resulted in death. Only the event that was
- 1322 the cause of death should be reported as fatal. AEs/SAEs that were ongoing at the time of death;
- however, were not the cause of death, will be recorded as "resolved" at the time of death. 1323
- 1324 NOT RECOVERED/NOT RESOLVED (ONGOING) - An ongoing AE/SAE is defined as the
- event was ongoing with an undetermined outcome. 1325
- 1326 o An ongoing outcome will require follow-up by the site in order to determine the final 1327 outcome of the AE/SAE.
- 1328 The outcome of an ongoing event at the time of death that was not the cause of death, 1329 will be updated and recorded as "resolved" with the date of death recorded as the stop 1330 date.
- 1331 UNKNOWN - An unknown outcome is defined as an inability to access the participant or the
- 1332 participant's records to determine the outcome (for example, a participant that was lost to follow-
- 1333 up).
- 1334 If any reported adverse events are ongoing when a participant completes the study (or withdraws),
- 1335 adverse events classified as UADEs will be followed until they are either resolved, or have no
- 1336 prospect of improvement or change, even after the participant has completed all applicable study
- 1337 visits/contacts. For all other adverse events, data collection will end at the time the participant

- completes the study. Note: participants should continue to receive appropriate medical care for an
- adverse event after their participation in the study ends.

# 1340 **10.3 Reportable Device Issues**

- All UADEs and ADEs as defined in section 10.2.1 will be reported on both a device issue form
- and AE form, except for skin reactions from CGM sensor placement or pump infusion set
- placement that do not require pharmacologic treatment. As noted in section 10.2.1, events that
- occur due to participant (user) error generally will not require completion of a device issue form.
- Such 'errors' could include improper use of an insulin pump or using a pump infusion set or
- 1346 CGM sensor for a period of time longer than its labeling.
- Device complaints and device malfunctions will be reported except in the following
- circumstances. These occurrences are expected and will not be reported on a Device Issue Form
- assuming criteria for a UADE or ADE have not been met:
- 1350 CGM sensor lasting fewer days than expected per manufacturer
- 1351 CGM tape adherence issues
- Battery lifespan deficiency due to inadequate charging or extensive wireless communication
- 1353 Intermittent device component disconnections/communication failures not requiring system
- replacement or workaround/resolution not specified in user guide/manual.
- Device issues clearly addressed in the user guide manual that do not require additional
- 1356 troubleshooting

# 1357 **10.4 Timing of Event Reporting**

- SAEs possibly related to a study device or study participation and UADEs must be reported to
- the Coordinating Center within 24 hours of the site becoming aware of the event. This can occur
- via phone or email, or by completion of the online serious adverse event form and device issue
- form if applicable. If the form is not initially completed, it should be competed as soon as
- possible after there is sufficient information to evaluate the event. All other reportable ADEs and
- other reportable AEs should be submitted by completion on the online form within 7 days of the
- site becoming aware of the event.
- The Coordinating Center will notify all participating investigators of any adverse event that is
- serious, related, and unexpected. Notification will be made within 10 working days after the
- 1367 Coordinating Center becomes aware of the event.
- Each principal investigator is responsible for reporting serious study-related adverse events and
- abiding by any other reporting requirements specific to his/her Institutional Review Board or
- 1370 Ethics Committee. Sites must report all serious, related adverse events within seven calendar
- 1371 days.
- Upon receipt of a qualifying event, the Sponsor will investigate the event to determine if a
- 1373 UADE is confirmed, and if indicated, report the results of the investigation to all overseeing
- 1374 IRBs, and the FDA within 10 working days of the Sponsor becoming aware of the UADE per

- 1375 21CFR 812.46(b) (2). The Medical Monitor must determine if the UADE presents an
- unreasonable risk to participants. If so, the Medical Monitor must ensure that all investigations,
- or parts of investigations presenting that risk, are terminated as soon as possible but no later than
- 1378 5 working days after the Medical Monitor makes this determination and no later than 15 working
- days after first receipt notice of the UADE.
- Device malfunctions will be handled by the Sponsor or designee as described below. In the case
- of a CGM transmitter or sensor device malfunction, information will be forwarded to Dexcom by
- the site personnel, to be handled by their complaint management system.

#### 1383 **10.5 Safety Oversight**

- 1384 The study Medical Monitor will review all adverse events and adverse device events that are
- reported during the study. SAEs typically will be reviewed within 24 hours of reporting. Other
- AEs typically will be reviewed on a weekly basis. Additionally, the Medical Monitor will review
- compiled safety data at periodic intervals (generally timed to the review of compiled safety data
- by the DSMB).
- 1389 The Protocol Chair will be informed of all cases of severe hypoglycemia and DKA and the
- Medical Monitor's assessment of relationship to the study device; and informed of all reported
- device issues.
- 1392 A Data and Safety Monitoring Board (DSMB) will be informed of all cases of severe
- 1393 hypoglycemia and diabetic ketoacidosis irrespective of device relationship, all device-related
- SAEs, and all UADEs at the time that they occur during the study and will review compiled
- safety data at periodic intervals. The DSMB also will be informed of any ADEs not meeting
- criteria for a UADE if the Medical Monitor requests the DSMB review. The DSMB can request
- modifications to the study protocol or suspension or outright stoppage of the study if deemed
- necessary based on the totality of safety data available. Details regarding DSMB review will be
- documented in a separate DSMB document.

# 1400 **10.6 Stopping Criteria**

1401

#### 10.6.1 Participant Discontinuation of Study Device

- In the case of an unanticipated system malfunction resulting in a severe hypoglycemia or DKA
- event (or a malfunction that could have led to severe hypoglycemia or DKA), use of the study
- pump will be suspended while the problem is diagnosed. The UADE will be reported to the IRB,
- DSMB, and FDA. After assessment of the problem and any correction, use of the closed-loop
- functionality will not be restarted until approval is received from the IRB, DSMB, and FDA.
- 1407 In the absence of a device malfunction, use of the study pump by a participant will be
- discontinued if any of the following occur:
- 1409 The investigator believes it is unsafe for the participant to continue on the intervention. This could
- be due to the development of a new medical condition or worsening of an existing condition; or
- participant behavior contrary to the indications for use of the device that imposes on the
- 1412 participant's safety

- 1413 The participant's parent requests that the treatment be stopped
- 1414 Two distinct episodes of DKA as defined in section 10.2.4
- 1415 Two distinct severe hypoglycemia events as defined in section 10.2.3
- One episode of DKA as defined in section 10.2.4 and one severe hypoglycemia event as defined
- 1417 in section 10.2.3
- Each DKA or severe hypoglycemia event will be reviewed by the Medical Monitor and by the
- DSMB with respect to determination of cause and whether the occurrence of the event can be
- attributed to use of the Control-IQ closed-loop feature.
- 1421 An additional requirement for continued study pump use following a single DKA or severe
- 1422 hypoglycemia event will be that (1) the site investigator believes that the event is explainable,
- unlikely to recur, and that it is safe for the participant to continue to use the system and (2) the
- Medical Monitor and DSMB concur. If either the Medical Monitor or DSMB determines that the
- occurrence of the event indicates that it is not safe for the participant to continue to use the study
- pump, use will be discontinued.
- Even if the study device system is discontinued, the participant will be encouraged to remain in
- the study through the final study visit
- 1429 **10.6.2** Criteria for Suspending or Stopping Overall Study
- In the case of an unanticipated system malfunction resulting in a severe hypoglycemia or severe
- 1431 hyperglycemia event (as defined in section 10.2.4), use of the study pump will be suspended while
- the problem is diagnosed.
- In addition, study activities could be similarly suspended if the manufacturer of any constituent
- study device requires stoppage of device use for safety reasons (e.g. product recall). The affected
- study activities may resume if the underlying problem can be corrected by a protocol or system
- modification that will not invalidate the results obtained prior to suspension.
- 1437 The study Medical Monitor and DSMB will review all adverse events and adverse device events
- that are reported during the study. SH and DKA event review will occur for each such event on an
- expedited basis, and compiled safety data, including SH and DKA event rates, will be reviewed at
- approximately 6-month intervals. The DSMB will be provided with age-specific DKA and SH
- rates from the T1D Exchange registry for means of comparison. The Medical Monitor or DSMB
- may request suspension of study activities or stoppage of the study if deemed necessary based on
- the totality of safety data available.

| 1444 | Chapter 11: Miscellaneous Considerations |
|---|---|
| 1445 | 11.1 Drugs Used as Part of the Protocol |
| 1446<br>1447 | Participants will use lispro, aspart, or glusiline rapid-acting insulin prescribed by their personal physician. |
| 1448 | 11.2 Collection of Medical Conditions and Medications |
| 1449<br>1450<br>1451 | <u>Pre-Existing Condition:</u> Any medical condition that is either present at screening, a chronic disease, or a prior condition that could impact the participant's health during the course of the study (e.g., prior myocardial infarction or stroke). |
| 1452<br>1453<br>1454<br>1455<br>1456 | Medical Conditions during the study: In addition to conditions meeting the reporting requirements for an adverse event or device issue as described above, the following medical conditions should also be reported: (1) new diagnosis of a chronic disease (i.e., not present at the time of enrollment), and (2) any medical condition that could affect the participant's ability to carry out any aspect of the protocol or could affect an outcome assessment. |
| 1457<br>1458<br>1459<br>1460<br>1461<br>1462<br>1463 | Medications: All medication for the treatment of chronic pre-existing conditions, medical conditions (including medical conditions that do not require recording), and/or adverse events that the participant is currently taking at screening and during the course of the study should be recorded. Nutraceuticals and preventative treatment also should be recorded. Medications only taken as needed either can be recorded when prescribed or only recorded if used during the study. Glucagon for treatment of severe hypoglycemia will only be recorded if used during the study. |
| 1464 | 11.3 Prohibited Medications, Devices, Treatments, and Procedures |
| 1465<br>1466<br>1467 | Participants using glulisine at the time of enrollment will be asked to contact their personal physician to change their prescribed personal insulin to lispro or aspart for the duration of the trial in the case they are randomized to experimental arm. |
| 1468<br>1469<br>1470 | Treatment with any non-insulin glucose-lowering agent (including GLP-1 agonists, Symlin, DPP-4 inhibitors, SGLT-2 inhibitors, biguanides, sulfonylureas and naturaceuticals) will not be permitted. |
| 1471<br>1472<br>1473<br>1474 | The investigational study devices (t:slim X2 insulin pump, study CGM systems) must be removed before Magnetic Resonance Imaging (MRI), Computed Tomography (CT) or diathermy treatment. Participants may continue in the trial after temporarily discontinuing use if requiring one of the treatments above. |
| 1475 | 11.4 Precautionary Medications, Treatments, and Procedures |
| 1476 | Not applicable. |

Not applicable.

11.5 Prophylactic Medications, Treatments, and Procedures

1477

#### 1479 11.6 Rescue Medications, Treatments, and Procedures

- All participants will be required to have a commercially available glucagon (or glucagon analog)
- preparation for treatment as needed of severe hypoglycemia.

# 1482 11.7 Participant Compensation

Participant compensation will be specified in the informed consent form.

# 1484 11.8 Participant Withdrawal

- Participation in the study is voluntary, and a participant may withdraw at any time. For participants
- who withdraw, their data will be used up until the time of withdrawal.

#### 1487 11.9 Confidentiality

- 1488 For security and confidentiality purposes, participants will be assigned an identifier that will be
- used instead of their name. Protected health information gathered for this study will be shared
- with the coordinating center, the Jaeb Center for Health Research in Tampa, FL. De-identified
- participant information may also be provided to research sites involved in the study.

1493

1494

1495

1496

1501

1502

1503

1504

1505

1506

1507

1508

1509 1510

#### 12.1 Statistical and Analytical Plans

The approach to sample size and statistical analyses are summarized below. A detailed statistical analysis plan will be written and finalized prior to the completion of the study.

# 12.2 Statistical Hypotheses

The primary outcome for this study is CGM-measured % in range 70-180 mg/dL over a 13-week period. The intervention will be considered effective if the Closed-Loop Control [CLC] is superior to Standard Care [SC] using a statistical significance of  $\alpha$ =0.05 and the model specified below in Section 6 (i.e., p < 0.05).

The null/alternative hypotheses are:

- a. *Null Hypothesis*: There is no difference in mean CGM-measured % in range 70-180 mg/dL over 13 weeks between SC and CLC
- b. *Alternative Hypothesis*: The mean CGM-measured % in range 70-180 mg/dL over 13 weeks is different for SC and CLC.

#### 12.3 Sample Size

Based on data from the DCLP5 study mentioned above, we conservatively estimate the standard deviation (SD) for the primary outcome, time in range (TIR), to be 10%. A sample size of N=90 subjects (60 in the CLC arm and 30 in the SC arm) therefore will give 90% power to detect a 7.5% improvement in TIR with a two-sided test and type 1 error of 5%. Accounting for potential attrition rate of up to 10%, the total sample size for the PEDAP Study is estimated at  $\underline{N=102}$ .

15111512

1513

1514

The following table shows the minimum detectable difference with a total sample size N=90 for key secondary outcomes. The observed standard deviations are taken from the DCLP5 study.

| | Standard Deviation | | | Correlation | | Detectable |
|---|---|---|---|---|---|---|
| Outcome | CLC<br>(n=78) | SC<br>(N=22) | Pooled<br>(N=100) | with<br>Baseline | Effective<br>SD <sup>a</sup> | Difference<br>with N=90 b |
| $\%$ >250 mg/dL $^{\rm c}$ | 5.5% | 9.9% | 6.5% | 0.69 | 4.7% | 3.4% |
| Mean Glucose d | 18 | 26 | 20 | 0.68 | 14 | 10 |
| HbA1c | 0.8% | 0.9% | 0.8% | 0.70 | 0.6% | 0.4% |
| $\%$ <70 mg/dL $^{\rm c}$ | 1.07% | 1.13% | 1.08% | 0.61 | 0.86% | 0.63% |
| % <54 mg/dL ° | 0.23% | 0.23% | 0.23% | 0.54 | 0.19% | 0.14% |

a – After accounting for the baseline value as a covariate in the regression model.

<sup>1516</sup> b – With 90% power and two-sided type 1 error rate = 5%.

<sup>1517</sup> c – Outcomes with a skewed distribution winsorized at the 10<sup>th</sup> and 90<sup>th</sup> percentiles.

<sup>1518</sup> d – Units for mean glucose are mg/dL.

- 1519 **12.4 Efficacy Outcome Measures**
- 1520 **12.4.1 Primary Efficacy Endpoint**
- CGM-measured % in range 70-180 mg/dL
- 1522 **12.4.2 Secondary Efficacy Endpoints**
- 1523 12.4.2.1 Secondary Efficacy Endpoints Included in Hierarchical Analysis
- 1524 The following secondary endpoints will be tested in a hierarchical fashion as described in
- 1525 section 12.7.1.
- CGM-measured % above 250 mg/dL
- CGM-measured mean glucose
- 1528 HbA1c at 13 weeks
- CGM-measured % below 70 mg/dL
- CGM-measured % below 54 mg/dL
- 1531 12.4.2.2 Other Secondary Efficacy Endpoints
- 1532 The following endpoints are considered exploratory. Type 1 error for these endpoints will be
- 1533 controlled using the false discovery rate (FDR) instead of the familywise error rate (FWER).
- 1534 *CGM-Measured*:
- 1535 % above 180 mg/dL
- 1536 % in range 70-140 mg/dL
- glucose variability measured with the coefficient of variation (CV)
- glucose variability measured with the standard deviation (SD)
- 1539 % <60 mg/dL
- low blood glucose index (LBGI)\*
- hypoglycemic events (defined as at least 15 consecutive minutes <54 mg/dL)
- hyperglycemic events (defined as at least 90 consecutive minutes >300 mg/dL)
- 1543 % > 300 mg/dL
- high blood glucose index (HBGI)\*
- % in range 70-180 mg/dL improvement from baseline to 13 weeks ≥5%
- % in range 70-180 mg/dL improvement from baseline to 13 weeks ≥10%
- % time in range 70-180 mg/dL >70% and % time <70 mg/dL <4%
- 1548 *HbA1c*:
- 1549 HbA1c < 7.0% at 13 weeks
- 1550 HbA1c < 7.5% at 13 weeks
- HbA1c improvement from baseline to 13 weeks >0.5%
- HbA1c improvement from baseline to 13 weeks >1.0%
- HbA1c relative improvement from baseline to 13 weeks >10%

1554 HbA1c absolute improvement from baseline to 13 weeks >1.0% or HbA1c <7.0% at 13 1555 weeks 1556 **Questionnaires** 1557 • PedsQL Diabetes Module – total score and 5 subscales: 1558 Diabetes 1559 o Treatment I 1560 o Treatment II 1561 Worry 1562 Communication 1563 Pediatric Inventory for Parents (PIP) 2 domains each with a total score and 4 subscales for (5x2=10 difference scores)1564 Frequency 1565 **Total Score** 1566 • 1567 Communication 1568 Medical Care 1569 **Role Function** 1570 Emotional Functioning 1571 o Difficulty Same total + 4 subscales as above for Frequency 1572 1573 • INSPIRE (CLC arm only) Pittsburgh Sleep Quality Index (PSQI) global score 1574 1575 Fear of Hypoglycemia Survey for Parents (HFS-P) – total score, 2 subscales and 4 factor 1576 scores: 1577 o Behavior 1578 Avoidance 1579 Maintain high BG 1580 Worry 1581 Helplessness 1582 Social consequences 1583 1584 \*Note that LBGI and HBGI will be calculated using all available CGM readings as described below. Therefore, they may not be comparable to the same metrics calculated with SMBG data. 1585 1586 Other: 1587 Insulin 1588 ♦ Total daily insulin (units/kg) 1589 ♦ Percentage of total insulin delivered via basal Weight and Body Mass Index (BMI) 1590 1591 12.4.3 CGM Metrics Calculations 1592 Randomization is preceded by 2-6 weeks of CGM run-in, which will be used in the calculation

of baseline CGM metrics. For participants who are eligible to skip the run-in, comparable

- amount of CGM data from their own sensors will be taken before randomization visit to
- 1595 calculate baseline CGM metrics.
- 1596 CGM data starting from randomization visit through the 13-week visit will be included in the
- 1597 calculation of each CGM metric. Percentages in range 70-180 mg/dL (and all other CGM-based
- metrics) will be calculated giving equal weight to each CGM point for each participant.

#### 1599 **12.5** Analysis Datasets and Sensitivity Analyses

- All analyses comparing the CLC arm with SC arm will follow intention-to-treatment approach,
- which means participants will be analyzed in the treatment arm assigned by randomization
- regardless of actual system use. All randomized participants will be included in the primary
- analysis and secondary hierarchical analyses of CGM metrics. For other secondary outcomes,
- only participants with non-missing outcome data will be included.
- Safety outcomes will be reported for all enrolled participants, irrespective of whether the
- participant was randomized or the study was completed.

# 1607 **12.5.1 Per Protocol Analyses**

- Per-protocol analyses will be performed for primary outcome and secondary hierarchical
- outcomes only if >5% of participants will be excluded:
- CLC arm: Closed loop mode active for at least 80% of the time
- SC arm: CGM use for at least 80% of the time

#### 1612 **12.5.2 Other Sensitivity Analyses**

- 1613 Confounding
- 1614 A sensitivity analysis will also be conducted if potential confounding factors collected at
- baseline are detected.
- 1616 The imbalance will be assessed based on clinical judgement reviewing the distributions in the
- two treatment arms, not on a p-value. The person making this judgement will be unaware of
- whether there is an association between baseline variables and study outcome. All variables
- obtained on a continuous scale will be entered into the models as continuous variables, unless it
- is determined that a variable does not have a linear relationship with the outcome. In such a case,
- 1621 categorization and/or transformation will be explored.
- 1622 Exclude First 2 Weeks of CGM Data
- The primary analysis will be repeated by excluding the first 2 weeks of post-randomization CGM
- 1624 data.
- 1625 Missing Data
- 1626 Missing data will be handled using direct likelihood method for the primary analysis. It is worth
- noting that all statistical methods for handling missing data rely on untestable assumptions and

- there is no one correct way to handle missing data. Our goal is to minimize the amount of
- missing data so that the results will not be sensitive to which statistical method is used.
- To that end, sensitivity analyses will be performed to explore whether results are similar for
- primary analysis when using different methods. The following methods will be applied:
- Rubin's multiple imputation with treatment group in the imputation model
- Available cases only
- Multiple imputation with pattern mixture model assuming the dropout trajectory of the
- 1635 CLC group was that of the SC group (Mallinckrodt and Clark, 2003) (3)

# 12.6 Analysis of the Primary Efficacy Endpoint

- Summary statistics (mean  $\pm$  SD or median (quartiles)) will be reported by treatment group for the
- 1638 CGM-measured % in range 70-180 mg/dL at baseline, 13 weeks intervention and change from
- baseline to 13 weeks.

1636

1661

- 1640 CGM-measured % in range 70-180 mg/dL between two treatment arms will be compared using a
- linear mixed effects regression model while adjusting for baseline CGM-measured % in range
- 1642 70-180 mg/dL, age, prior CGM and pump use, and clinical center (random effect). A point
- estimate, 95% confidence interval and two-sided p-value will be reported for the treatment effect
- based on the linear regression model and a 5% level will be used to declare statistical
- significance. Residual values will be examined for an approximate normal distribution. If values
- are highly skewed then robust regression using M-estimation will be used instead. However,
- previous experience suggests that the residual values for % time glucose in target range will
- follow an approximately normal distribution. Imbalances between groups in important covariates
- are not expected to be of sufficient magnitude to produce confounding. However, the presence of
- 1650 confounding will be evaluated in the sensitivity analyses by including factors potentially
- associated with the outcome for which there is an imbalance between groups (12.5.2).
- In the primary analysis, any missing data at baseline or follow-up will be handled using direct
- likelihood. A longitudinal linear regression model will be fit with the percent of time in range at
- baseline and follow-up as the dependent variable. This model will adjust for age, prior CGM use
- and pump use as fixed effects and clinical center as a random effect. This model adjusts for
- baseline time in range by forcing the treatment groups to have the same mean value at baseline.

#### 1657 **12.7** Analysis of the Secondary Endpoints

- Point estimates and confidence intervals for the treatment arm differences will be presented for
- all secondary metrics. The models will adjust for the corresponding baseline metric, age, prior
- 1660 CGM and pump use, and clinical center (random effect).

#### 12.7.1 Hierarchical Analyses

- To preserve the overall type 1 error for selected key secondary endpoints, a hierarchical testing
- procedure will be used. If the primary analysis for time in range described above results in a
- statistically significant result (p < 0.05), then testing (similar to the model described above
- 1665 for the primary outcome) will proceed to the next outcome metric in the following order:

- CGM-measured % in range 70-180 mg/dL (primary outcome)
- CGM-measured % above 250 mg/dL
- CGM-measured mean glucose
- HbA1c at 13 weeks
- CGM-measured % below 70 mg/dL
- CGM-measured % below 54 mg/dL

1672

- 1673 This process continues iteratively moving to the next variable down on the list until a non-
- significant result ( $p \ge 0.05$ ) is observed, or all six variables have been tested. If a non-significant
- result is encountered, then formal statistical hypothesis testing is terminated and any variables
- below on the list are not formally tested.
- Regardless of the results of the hierarchical testing, summary statistics appropriate to the
- distribution will be tabulated by treatment arm for each hierarchical outcome. A 95% confidence
- interval for the treatment arm difference will also be calculated for all five secondary hierarchical
- outcomes listed above. However, a confidence interval that excludes zero will not be considered
- a statistically significant result if an outcome variable higher on the hierarchical list failed to
- reach statistical significance.
- Analysis for each of the CGM metrics listed above for the hierarchical analysis will parallel the
- analysis described for the primary outcome in Section 12.6.
- HbA1c at 13 weeks will be compared between the two treatment arms using a linear model while
- adjusting for baseline HbA1c, age, prior CGM and pump use, and clinical center (random
- factor). Missing data will be handled using direct likelihood in a regression model including all
- available central laboratory HbA1c measurements at baseline and 13-week visits.
- 1689 For all above analyses, regression diagnostics will be employed analogous to as described in
- 1690 Section 12.6 for the primary outcome.

#### 1691 **12.7.2 Other Endpoint Analyses**

- 1692 For all other secondary endpoints, only participants with non-missing data will be included in
- analyses (available cases method). Summary statistics (mean  $\pm$  SD, median (IQR) or n (%))
- appropriate to the distribution will be tabulated for them at baseline, 13 weeks and for the
- 1695 changes from baseline to 13 weeks. For continuous outcomes, linear regression models will be
- used to compare the treatment effects while adjusting for corresponding baseline values (e.g.,
- baseline % in range 70-140 mg/dL for comparing change in % in range 70-140 mg/dL from pre-
- randomization CGM wear to 13 weeks post-randomization period), age, prior CGM and pump
- use, and clinical center as a random effect. Comparisons of body weight and BMI will also be
- adjusted for gender.
- For CGM-measured hypoglycemia/hyperglycemia events, event rates per week will be compared
- using similar linear mixed effects regression models as described above for the primary outcome.

1703

#### 1704 Binary HbA1c and CGM Outcomes

- 1705 For the binary HbA1c outcomes, risk-adjusted percentages by treatment group will be computed
- at 13 weeks from a logistic regression model. The logistic regression will adjust for baseline
- HbA1c (as a continuous factor), age, prior CGM and pump use as fixed effects, and clinical site
- as a random effect. Similar analyses will be done for the binary CGM outcomes.

#### 1709 *Questionnaires*

- For each questionnaire, mean  $\pm$  SD or percentiles appropriate to the distribution will be given by
- treatment group at baseline and 13 weeks. Group comparisons will be conducted for the total
- score (mean score) and subscales from participant version and parent version separately using
- similar linear models as described above. The INSPIRE and SUS post-treatment surveys will
- only be administered to the CLC group at the 13-week visit, and thus the scores will only be
- 1715 tabulated.

#### 1716 Focus Groups

- 1717 Qualitative data from focus groups will be analyzed using NVIVO (release 11.2; QSR
- 1718 International) to organize and manage the entire corpus of focus group data. Analysis begins
- with an initial coding procedure to capture and describe the range of responses to the
- intervention. A second, more focused and detailed level of coding will be applied to major
- categories of findings in the initial review to determine themes in response to the clinical trial,
- use of the closed loop system, and quality of life changes. The video data from the co-regulation
- interaction will be submitted to the validated coding system and frequencies of positive and
- 1724 negative interactions, treatment discussions, and CLC comments will be calculated with simple
- descriptive statistics. Change from pre to post treatment will be analyzed in the similar GLM
- framework to evaluate whether there is improvement in co-regulation across the study.
- 1727 Boxplots
- Boxplots stratified by treatment group will be given for the primary outcome and each of the key
- secondary endpoints in specified time periods over the 13-week course of follow-up.

#### 1730 12.8 Safety Analyses

- All randomized participants will be included in these analyses and all their post-randomization
- safety events will be reported. Any pre-randomization adverse events will be tabulated separately
- and will include any participants who were never randomized.
- Safety analyses of the main study (randomized trial phase) will include events occurring on or
- after randomization until and including the 13-week visit or Day 105 from randomization,
- 1736 whichever occurs first. Safety analyses of the extension phase will include subsequent events
- until the last visit date or the last event date (whichever is later).
- 1738 For the following outcomes, the number of events will be tabulated by treatment group. Formal
- statistical comparisons (main study phase only) will be performed if there are enough events (at
- least 5 events combined between the two treatment groups):
- Number of SH events and SH event rate per 100 person-years

- Number of DKA events and DKA event rate per 100 person-years
- Other serious adverse events
- Any adverse event rate
- Number of calendar days with any ketone level ≥1.0 mmol/L (if ≥5 total calendar days combined)
- Worsening of HbA1c from baseline to 13 weeks by >0.5%
- Investigational device related (intervention group only):
- 1749 Adverse device effects (ADE)
- o Serious adverse device events (SADE)
- 1751 o Unanticipated adverse device effects (UADE)

1752

- 1753 For DKA and SH events, if enough events, the rates will be compared between the two treatment
- arms during the main study phase using a robust Poisson regression. The regression will adjust
- for the participant-reported number of SH events 12 months prior to the start of the study and
- clinical center as random effect. The amount of follow up will be included as an offset covariate
- to compare the rates. A similar analysis will be done for DKA, if at least 5 total DKA events
- among both treatment groups.

1759

1760

#### 12.9 Intervention Adherence

- 1761 The following tabulations and analyses will be performed by treatment group to assess
- intervention adherence for the study:
- Sensor use –percent time of use, overall for 13-week visit
- 1764 For CLC arm only, the following will be tabulated to assess adherence:
- Closed loop system use–percent time of use, overall for 13-week visit
- % time in different operational modes overall and by specified time periods

#### 1767 **12.10 Protocol Adherence and Retention**

- 1768 The following tabulations and analyses will be performed by treatment group to assess protocol
- adherence for the study:
- Number of protocol and procedural deviations
- Flow chart accounting for all enrolled participants up to randomization
- Flow chart of all randomized participants at all scheduled visits and phone contacts post
- treatment initiation
- Number of and reasons for unscheduled visits and phone calls
- Number of participants who stopped treatment and reasons

#### 1776 **12.11 Baseline Descriptive Statistics**

- Baseline demographic and clinical characteristics of the cohort of all randomized participants
- will be summarized in a table using summary statistics appropriate to the distribution of each
- variable. Descriptive statistics will be displayed by treatment group for the following:

- 1780 Age
- 1781 Sex
- 1782 Race/Ethnicity
- Parent's income, education, and/or insurance status
- 1784 Diabetes duration
- Insulin method before enrollment (pump vs. MDI)
- CGM use before enrollment
- 1787 HbA1c
- 1788 BMI %
- Participant-reported number of SH and DKA 12 months prior to the start of the study
- Baseline CGM metrics including:
- % in range 70-180 mg/dL
- 1792 % time > 180 mg/dL
- Mean glucose
- % time < 70 mg/dL
- 1795 % time < 54 mg/dL

#### 1796 **12.12 Device Issues**

- 1797 The following tabulations and analyses will be performed by treatment group to assess device
- 1798 issues:
- Device malfunctions requiring study team contact and other reported device issues
- Rate of different failure events and alarms per 24 hours recorded by the Control-IQ system overall and by month

#### 1802 **12.13 Planned Interim Analyses**

- No formal interim efficacy analyses are planned. The analysis of the RCT will be performed on
- 1804 completion of the RCT prior to the completion of the extension phase.
- In addition, the DSMB will review safety data at intervals, with no formal stopping rules.

#### 1806 **12.14 Subgroup Analyses**

- In exploratory analyses, the primary outcome (time 70-180 mg/dL), % time <70 mg/dL and HbA1c
- at 13 weeks will be assessed separately in various subgroups. Subgroups will be defined according
- 1809 to the baseline value of the factors, which will be noted in the SAP. Tests for interaction
- 1810 with treatment group will be performed.
- 1811 Interpretation of subgroup analyses will be viewed with caution, particularly in the absence of an
- overall significant difference. For continuous variables, results will be displayed in subgroups
- based on cutpoints although the analysis will utilize the variable as continuous. If there is
- 1814 insufficient sample size in a given subgroup, the cutpoints for continuous measures may be
- adjusted per the observed distribution of values. Cutpoint selection for display purposes will be
- 1816 made masked to the outcome data.
#### 1817 12.15 Multiple Comparison/Multiplicity 1818 Primary Analysis 1819 Since there will be a single comparison for the primary outcome (CGM-measured % 70-180 1820 mg/dL), no adjustment is needed. 1821 Secondary Hierarchical Analyses 1822 The hierarchical testing procedure described above in section 12.7.1 will be used to control the overall type 1 error for the primary outcome plus five key secondary outcomes identified above. 1823 1824 All Other Secondary Analyses 1825 For comparison of all other efficacy endpoints, the false discovery rate will be controlled using the 1826 adaptive Benjamini-Hochberg procedure (4). 1827 P-values from safety analyses, sensitivity analyses, and per-protocol analyses will not be adjusted 1828 for multiple comparisons. 1829 12.16 Exploratory Analyses 1830 CGM Metrics 1831 In addition to the analysis for the CGM-measured endpoints described earlier, separate analyses 1832 will be conducted for daytime and nighttime of the following metrics: • % time in range 70-180 mg/dL 1833 1834 • Mean glucose • % above 180 mg/dL 1835 % below 70 mg/dL 1836 coefficient of variation 1837 1838 1839

- Above selected CGM metrics also will be reported by restricting the CGM data in the CLC arm based on following criteria. No p-values will be calculated for following analyses.
  - using only the CGM data when the closed-loop is active

1841 1842

- 1843 Additional Insulin Metrics
- The following insulin metrics will be tabulated by treatment groups at baseline, 13 weeks and for the changes from baseline to 13 weeks. No p-values will be calculated for these metrics.
- Total daily basal insulin (units/kg)
  - Total daily bolus insulin (units/kg)
  - Total daily manual bolus (units/kg)
- Total daily automated bolus (units/kg)
- Total daily short-acting injections for injection users

1851

1847

- The following will be calculated for the CLC group in the 1-week prior to randomization and by 1-week follow-up periods from pump data only:
- Total daily insulin (units/kg)
- Total daily basal insulin (units/kg)
- Total daily bolus insulin (units/kg)
  - o Total daily manual bolus (units/kg)
- 1858 Total daily automated bolus (units/kg)
- Number of manual insulin doses per day
- Number of manual insulin doses with carb announcement per day

1861

1862

1857

#### 12.17 Extension Phase

Analyses for the extension phase will be primarily exploratory.

1864

- For both treatment arms, summary statistics will be given for all outcomes listed above in
- Section 12.4 at RCT baseline (pre-randomization), 13 weeks, and 26 weeks. In addition, boxplots
- will be constructed for each of the outcome metrics listed above showing both treatment arms
- over the course of the combined RCT and extension (where both arms using CLC) phases.
- Formal statistical comparisons between the two study phases (i.e., primary RCT and extension
- phases) will be performed for key outcome measures including:
- CGM-measured % in range 70-180 mg/dL
- CGM-measured % above 250 mg/dL
- CGM-measured mean glucose
- 1874 HbA1c at 13 weeks
- CGM-measured % below 70 mg/dL
- CGM-measured % below 54 mg/dL
- PedsOL Diabetes Module total score
- Pediatric Inventory for Parents (PIP)
- Frequency domain total score
  - ➤ Difficulty domain total score
- 1881 INSPIRE Survey
- Pittsburgh Sleep Quality Index (PSQI) global score
- Fear of Hypoglycemia Survey for Parents (HFS-P) total score
- Hypoglycemia Confidence Scale (HCS)
- System Usability Scale (SUS)
- For each of these outcomes a longitudinal regression model will be fit combining data from the
- 1887 RCT and extension phases accounting for the correlated data from repeated measures. Treatment
- group will be a time dependent factor in this model. A point estimate and 95% confidence
- interval will be given for the estimated effects of each CLC version used during the study, both
- with respect to SC and with respect to one another. Safety analyses of the Extension Phase will
- include events occurring on or after the Extension training visit until the end of the 26-Week visit

1893 outcomes will include those specified in section 12.8 with the exception of worsening of HbA1c. 1894 Summary statistics appropriate to the distribution will be tabulated without any formal 1895 comparisons by treatment group for the safety outcomes noted in section 12.8. 1896 12.17.1 Exclusion of Ancillary Study Data 1897 According to Chapter 14, during the extension phase, 30-40 participants will be sought to enroll in an ancillary study to test the Control-IQ system with meal bolus and exercise 1898 challenges. The analyses for this ancillary study are specified in Section 14.5. Data collected 1899 1900 from the start of each of these challenges until 5:59 AM the following morning will be excluded from the analysis of the extension phase. 1901 1902 1903 12.18 Extended Use Period 1904 Analyses for the extended use phase will be exploratory. 1905 1906 Summary statistics will be given for all outcomes listed above in Section 12.4 for each of the 13-1907 week periods following initiation of the Extended Use period. In addition, boxplots will be 1908 constructed for each of the outcome metrics listed above for these periods. 1909 1910 Safety analyses of the Extended Use period will include events until the last visit date or the last 1911 event date (whichever is later). Safety outcomes will include those specified in section 12.8 with 1912 the exception of worsening of HbA1c. 1913

or the end of Day 105 from the Extension training visit — whichever occurs first. Safety

# **Chapter 13: Data Collection and Monitoring**

| 1915 | 13.1 Case Report Forms and Device Data |
|---|---|
| 1916<br>1917<br>1918<br>1919<br>1920<br>1921<br>1922<br>1923 | The main study data are collected on electronic case report forms (CRFs). When data are directly collected in electronic case report forms, this will be considered the source data. For any data points for which the eCRF is not considered source (e.g. lab results that are transcribed from a printed report into the eCRF), the original source documentation must be maintained in the participant's study chart or medical record. This source must be readily verifiable against the values entered into eCRF. Even where all study data are directly entered into the eCRFs at office visits, evidence of interaction with a live subject must be recorded (e.g., office note, visit record, etc.). |
| 1924<br>1925 | Electronic device data files are obtained from the study software and individual hardware components. These electronic device files are considered the primary source documentation. |
| 1926 | 13.2 Study Records Retention |
| 1927<br>1928<br>1929 | Each participating site will maintain appropriate medical and research records for this trial, in compliance with ICH E6 and regulatory and institutional requirements for the protection of confidentiality of participants. |
| 1930<br>1931<br>1932<br>1933<br>1934<br>1935<br>1936 | Study documents should be retained for a minimum of 2 years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or until at least 2 years have elapsed since the formal discontinuation of clinical development of the investigational product. These documents should be retained for a longer period, however, if required by local regulations. No records will be destroyed without the written consent of the sponsor, if applicable. It is the responsibility of the sponsor to inform the investigator when these documents no longer need to be retained. |
| 1937 | 13.3 Quality Assurance and Monitoring |
| 1938<br>1939<br>1940<br>1941<br>1942<br>1943 | Designated personnel from the Coordinating Center will be responsible for maintaining quality assurance (QA) and quality control (QC) systems to ensure that the clinical portion of the trial is conducted and data are generated, documented and reported in compliance with the protocol, Good Clinical Practice (GCP) and the applicable regulatory requirements, as well as to ensure that the rights and wellbeing of trial participants are protected and that the reported trial data are accurate, complete, and verifiable. Adverse events will be prioritized for monitoring. |
| 1944<br>1945<br>1946<br>1947<br>1948 | A risk-based monitoring (RBM) plan will be developed and revised as needed during the course of the study, consistent with the FDA "Guidance for Industry Oversight of Clinical Investigations — A Risk-Based Approach to Monitoring" (August 2013). Study conduct and monitoring will conform with 21 Code of Federal Regulations (CFR) 812. This plan describes in detail who will conduct the monitoring, at what frequency monitoring will be done, at what level of detail monitoring will be performed, and the distribution of monitoring reports. |

- 1950 The data of most importance for monitoring at the site are participant eligibility and adverse
- events. Therefore, the RBM plan will focus on these areas. As much as possible, remote
- monitoring will be performed in real-time with on-site monitoring performed to evaluate the
- verity and completeness of the key site data. Elements of the RBM may include:
- Qualification assessment, training, and certification for sites and site personnel
- Oversight of Institutional Review Board (IRB) coverage and informed consent procedures
- Central (remote) data monitoring: validation of data entry, data edits/audit trail, protocol review of entered data and edits, statistical monitoring, study closeout
- On-site monitoring (site visits): source data verification, site visit report
- Agent/Device accountability
- Communications with site staff
- Patient retention and visit completion
- Quality control reports
- Management of noncompliance
- Documenting monitoring activities
- Adverse event reporting and monitoring
- 1966 Coordinating Center representatives or their designees may visit the study facilities at any time in
- order to maintain current and personal knowledge of the study through review of the records,
- comparison with source documents, observation and discussion of the conduct and progress of the
- 1969 study. The investigational site will provide direct access to all trial related sites, source
- data/documents, and reports for the purpose of monitoring and auditing by the sponsor, and
- inspection by local and regulatory authorities.
- 1972 **13.4 Protocol Deviations**
- 1973 A protocol deviation is any noncompliance with the clinical trial protocol, GCP, or procedure
- requirements. The noncompliance may be either on the part of the participant, the investigator,
- or the study site staff. As a result of deviations, corrective actions are to be developed by the site
- and implemented promptly.
- 1977 The site PI/study staff is responsible for knowing and adhering to their IRB requirements. Further
- details about the handling of protocol deviations will be included in the monitoring plan.

## **Chapter 14: Ethics/Protection of Human Participants**

#### 1980 14.1 Ethical Standard

1979

1984

1991

1992

2009

- 1981 The investigator will ensure that this study is conducted in full conformity with Regulations for
- the Protection of Human Participants of Research codified in 45 CFR Part 46, 21 CFR Part 50, 21
- 1983 CFR Part 56, and/or the ICH E6.

#### 14.2 Institutional Review Boards

- 1985 The protocol, informed consent form(s), recruitment materials, and all participant materials will
- be submitted to the IRB for review and approval. Approval of both the protocol and the consent
- 1987 form must be obtained before any participant is enrolled. Any amendment to the protocol will
- require review and approval by the IRB before the changes are implemented to the study. All
- changes to the consent form will be IRB approved; a determination will be made regarding whether
- previously consented participants need to be re-consented.

#### 14.3 Informed Consent Process

### 14.3.1 Consent Procedures and Documentation

- 1993 Informed consent is a process that is initiated prior to the individual's agreeing to participate in
- the study and continues throughout the individual's study participation. Extensive discussion of
- risks and possible benefits of participation will be provided to the participants and their families.
- 1996 Consent forms will be IRB-approved and the participant will be asked to read and review the
- document. The investigator will explain the research study to the participant and answer any
- 1998 questions that may arise. All participants will receive a verbal explanation in terms suited to
- their comprehension of the purposes, procedures, and potential risks of the study and of their
- 2000 rights as research participants. Participants will have the opportunity to carefully review the
- written consent form and ask questions prior to signing.
- The participants should have the opportunity to discuss the study with their surrogates or think
- about it prior to agreeing to participate. The participant will sign the informed consent document
- prior to any procedures being done specifically for the study. The participants may withdraw
- 2005 consent at any time throughout the course of the trial. A copy of the informed consent document
- will be given to the participants for their records. The rights and welfare of the participants will
- be protected by emphasizing to them that the quality of their medical care will not be adversely
- affected if they decline to participate in this study.

#### 14.3.2 Participant and Data Confidentiality

- 2010 Participant confidentiality is strictly held in trust by the participating investigators, their staff,
- and the sponsor(s) and their agents. This confidentiality is extended to cover testing of
- 2012 biological samples and genetic tests in addition to the clinical information relating to
- 2013 participants. Therefore, the study protocol, documentation, data, and all other information
- 2014 generated will be held in strict confidence. No information concerning the study or the data will
- be released to any unauthorized third party without prior written approval of the sponsor.

2016 The study monitor, other authorized representatives of the sponsor, representatives of the IRB, 2017 regulatory agencies or company supplying study product may inspect all documents and records 2018 required to be maintained by the investigator, including but not limited to, medical records 2019 (office, clinic, or hospital) and pharmacy records for the participants in this study. The clinical 2020 study site will permit access to such records. 2021 The study participant's contact information will be securely stored at each clinical site for internal use during the study. At the end of the study, all records will continue to be kept in a 2022 2023 secure location for as long a period as dictated by the reviewing IRB, institutional policies, or 2024 sponsor requirements. 2025 Study participant research data, which is for purposes of statistical analysis and scientific reporting, 2026 will be transmitted to and stored at the Jaeb Center for Health Research (JCHR). This will not 2027 include the participant's contact or identifying information, unless otherwise specified in the 2028 informed consent form. Rather, individual participants and their research data will be identified 2029 by a unique study identification number. The study data entry and study management systems 2030 used by clinical sites and by JCHR research staff will be secured and password protected. At the 2031 end of the study, all study databases will be de-identified and archived at the JCHR and the 2032 University of Virginia Center for Diabetes Technology.

| 2034 | <b>Chapter 15: Ancillary Study to Test Control-IQ System with Meal</b> |
|---|---|
| 2035 | <b>Bolus and Exercise Challenges</b> |
| 2036 | 15.1 Objective |
| 2037<br>2038<br>2039 | This Ancillary Study will assess the safety of using the study system during exercise and meal bolus-related challenges. Outcome data are expected to be used to support regulatory filings for the device system. |
| 2040 | 15.2 Sample Size |
| 2041<br>2042<br>2043 | Participation in the Ancillary Study will be offered to participants who are currently in the Extension Phase of the main study. The goal for sample size is to have 30-40 individuals participate in the Ancillary Study. |
| 2044 | 15.3 Eligibility Criteria |
| 2045<br>2046<br>2047 | Participants must be currently in the Extension Phase of the main study, with at least 2 weeks and no more than 11 weeks completed to ensure sufficient comfort with the study pump and sufficient time to complete the protocol below. |
| 2048<br>2049 | Inclusion in the Ancillary Study requires investigator judgment that it is safe for the individual to participate. |
| 2050 | 15.4 Study Procedures |
| 2051<br>2052 | On the day of enrollment into the Ancillary Study, informed consent will be obtained from interested participants, and eligibility will be verified. |
| 2053<br>2054<br>2055 | A paper logbook will be provided to participants that includes a page to record details about each challenge and procedural instructions about how participants will conduct these challenges. This material will be reviewed with each participant. |
| 2056<br>2057<br>2058<br>2059<br>2060<br>2061 | During home use, each participant will perform 3 exercise and meal bolus-related challenges (details below) appropriate for the age of the participant. Each challenge will be separated from the other challenges by at least 48 hours. Before starting each challenge, caregivers of the child must assure the child has a working CGM and Control-IQ is active. If activity is paused during an exercise-related challenge, the challenge may be continued to allow for continuation of the activity if the participant is able and willing to continue. |
| 2062<br>2063 | Participants will receive a guidance document for performing the challenges that includes the following safety mitigations: |
| 2064<br>2065<br>2066 | • The participant's parent or guardian must remain with the child at all times and monitor CGM readings frequently during and for at least two hours after completion of each challenge. |

- The hyperglycemia safety protocol described in section 8.2.4 will be followed during each challenge.
  - The parent/guardian must have an on-call phone number for the study team prior to initiation of each challenge.
    - CGM glucose must be ≥120 mg/dL prior to initiation of each exercise-related challenge.
    - Exercise may not be initiated during an exercise-related challenge if the CGM trend arrows on the study insulin pump indicate Falling glucose (down arrow) or Rapidly Falling glucose (double down arrow).
    - Snacks and glucagon must be available for use during and after each exercise-related challenge.
    - Control-IQ exercise activity mode must be activated at least 30 minutes prior to the start of exercise during each exercise-related challenge and kept active for at least 30 minutes after completion of the exercise period.
    - Additional carbohydrate may be given as needed at the start of, during, or after each exercise-related challenge.
    - The temporary basal rate feature of the study pump may be used if desired to reduce insulin delivery during the exercise period of each exercise-related challenge.
    - Fingersticks will be performed for any low CGM value <70 mg/dL, and any exercise should be stopped if BG is confirmed <70 mg/dL. Exercise may be stopped for concerns for CGM decreasing at any time, even if CGM is >70 mg/dL.
    - A parent/guardian will sleep in the same home as the child overnight and closely monitor CGM readings following days when one of the challenges was performed.
- 2090 Contact with the study investigator may be initiated at any time.
- 2091 Challenge Details:
- 2092 Missed Meal Bolus Challenge: Participants will skip their meal bolus for an afternoon meal of
- at least 20 grams carbohydrate. The meal timing and carb amount and any additional snacks
- 2094 given will be recorded on a study exercise log. Additional insulin boluses may be given for
- 2095 hyperglycemia as needed. The hyperglycemia safety protocol described in section 8.2.4 will be
- 2096 followed.

2069

2070

2071 2072

2073

2074

2075

2076

2077

2078

2079

2080

2081

2082

2083

2084

2085

2086

2087

2088

- 2097 Full Meal Bolus Plus Exercise Challenge: Participants will receive a full meal bolus for an
- afternoon meal of at least 20 grams carbohydrate. The pump's Exercise Activity setting will be
- 2099 turned on upon completion of the meal. Beginning 30 minutes after completion of the meal, a
- 2100 parent/guardian will try to keep the child physically active (walking, running, playing) for at
- 2101 least 30 minutes if possible, or longer if desired. This can be mixed with mild activity. The meal
- 2102 timing and carb amount, the actual stop and start time of exercise, any associated hypoglycemia
- treatments, and any additional snacks given will be recorded on a study exercise log.

- 2104 **Exercise Challenge:** At least 2 hours after the child finishes an afternoon meal, a
- 2105 parent/guardian will try to keep the child physically active (walking, running, playing) for at
- least 30 minutes if possible, or longer if desired. This can be mixed with mild activity. The 2106
- 2107 pump's Exercise Activity setting will be turned on 90 minutes after completion of the meal. The
- meal timing and carb amount of the last meal prior to exercise, the actual start and stop time of 2108
- 2109 exercise, any associated hypoglycemia treatments, and any additional snacks given will be
- 2110 recorded on a study exercise log.
- 2111 A challenge may be stopped for any reason, including participant non-cooperation, or concern
- 2112 for hypoglycemia, or repeated hypoglycemia.
- 2113 15.5 Outcomes and Analysis Plan
- 2114 A separate statistical analysis plan will be written for the Ancillary Study.
- 2115 Outcomes will include the following:
- 2116 **Key Safety Outcomes:**
- 2117 Severe hypoglycemia
- 2118 • Other adverse events
- 2119 All adverse events will be listed. Listings will include Participant ID, the event, whether the
- 2120 event was serious, whether the event was related to the study device, the event outcome, and a
- 2121 description of the event.
- 2123 **Other Outcomes**

- 2124 CGM-measured % <54 mg/dL overnight (all challenge types)
- 2125 • CGM-measured % <70 mg/dL overnight (all challenge types)
- 2126 • CGM-measured % >180 mg/dL overnight (all challenge types)
- 2127 CGM-measured % <54 mg/dL during the two hours immediately following the start of exercise for each exercise-related challenge 2128
- 2129 • CGM-measured % <70 mg/dL during the two hours immediately following the start of 2130 exercise for each exercise-related challenge
- 2131 • CGM-measured % >180 mg/dL during the four hours following the announced meal, or 2132 until the next meal bolus is given, for the missed meal bolus challenge
- 2133 CGM-measured % >300 mg/dL during the four hours following the announced meal, or 2134 until the next meal bolus is given, for the missed meal bolus challenge
- 2135 The percentage of time spent below 54 mg/dL from 10 PM - 5.59 AM the night of an exercise
- 2136 challenge will be compared with percentage of time spent below 54 mg/dL the previous night
- using a linear mixed effects regression model. A point estimate, 95% confidence interval and 2137
- 2138 two-sided p-value will be reported for the challenge effect based on the linear regression model
- 2139 and a 5% level will be used to declare statistical significance. Residual values will be examined
- 2140 for an approximate normal distribution. If values are highly skewed, then robust regression using
- 2141 M-estimation will be used instead. Analysis of the percentage of time spent below 70 mg/dL 10

2142 PM – 5:59 AM the night of an exercise challenge will be performed in the same manner.

2143

- 2144 The percentage of time spent above 180 mg/dL from 10 PM - 5.59 AM the night of a missed
- meal bolus challenge will be compared with percentage of time spent above 180 mg/dL the 2145
- 2146 previous night using a linear mixed effects regression model. A point estimate, 95% confidence
- 2147 interval and two-sided p-value will be reported for the challenge effect based on the linear
- 2148 regression model and a 5% level will be used to declare statistical significance. Residual values
- will be examined for an approximate normal distribution. If values are highly skewed, then 2149
- 2150 robust regression using M-estimation will be used instead. Analysis of the percentage of time
- 2151 spent above 300 mg/dL 10 PM – 5:59 AM the night of a missed meal bolus challenge will be
- performed in the same manner. 2152

2153

- 2154 CGM-measured % <54 mg/dL during the two hours immediately following the start of exercise
- 2155 for each exercise challenge will be compared between the two exercise challenge groups using a
- 2156 paired t-test. CGM-measured % <70 mg/dL during this same period will be analyzed in the same
- 2157 manner.

- 2159 For each challenge type, the mean, standard deviation, and range will be given for the outcomes
- 2160 listed above relevant to the challenge type. Summary statistics for the overnight periods
- preceding the challenges will be presented with summary statistics for each challenge type. 2161
- 2162 **Safety Monitoring**
- 2163 Safety oversight will be the same as for the main study, as described in Chapter 10:.

## **Chapter 16: References**

- 2164
- 2165 1. Brown S, Kovatchev B, Raghinaru D, Lum JW, Buckingham BA, Kudva YC, Laffel LM,
- Levy CJ, Pinsker JE, Wadwa RP, Dassau E, Doyle FJ, Anderson SM, Church MM, Dadlani
- V, Ekhlaspour L, Forlenza GP, Isganaitis E, Lam DW, Kollman C, and Beck RW, for the
- 2168 iDCL Trial Research Group: Six-Month Randomized, Multicenter Trial of Closed-Loop
- 2169 Control in Type 1 Diabetes. N Engl J Med. 2019 Oct 31;381(18):1707-1717. doi:
- 2170 10.1056/NEJMoa1907863.
- 2171 2. Breton MD, Kanapka LG, Beck RW, Ekhlaspour L, Forlenza GP, Cengiz E, Schoelwer M,
- Ruedy KJ, Jost E, Carria L, Emory E, Hsu LJ, Oliveri M, Kollman CK, Dokken BB, Weinzimer
- SA, DeBoer MD, Buckingham BA, Cherñavvsky D, and Wadwa RP, for the iDCL Trial
- 2174 Research Group: A Randomized Trial of Closed-Loop Control in Children with Type 1
- 2175 Diabetes. N Engl J Med. 2020 Aug 27;383(9):836-845. doi: 10.1056/NEJMoa2004736.
- 3. Mallinckrodt CH, Clark WS, et al: Assessing responses profiles from incomplete longitudinal clinical trial data under regulatory considerations, J. Biopharm. Stat., 2003; 13(2): 179-190.
- 4. Benjamini, Y. and Hochberg, Y. (1995) Controlling the false discovery rate: a practical and powerful approach to multiple testing. J. R. Statist. Soc. B, 57, 289–300.